Study Protocol

Protocol Number: MT-1186-A04

A Phase 3b, Multicenter, Randomized, Double-blind

Extension Study to Evaluate the Continued Efficacy

and Safety of Oral Edaravone Administered for an

Additional Period of up to 48 Weeks Following Study

MT-1186-A02 in Subjects with Amyotrophic Lateral

Sclerosis (ALS)

Version Number: 3.0

Date: 29 July 2022

NCT number: NCT05151471

# STUDY PROTOCOL

**Protocol Number: MT-1186-A04** 

A Phase 3b, Multicenter, Randomized, Double-blind Extension Study to Evaluate the Continued Efficacy and Safety of Oral Edaravone Administered for an Additional Period of up to 48 Weeks Following Study MT-1186-A02 in Subjects with Amyotrophic Lateral Sclerosis (ALS)

IND Number:

138145

**EudraCT Number:** 

2021-003900-42

**Investigational Medicinal** 

Edaravone (MT-1186)

**Product:** 

Indication:

Treatment of Amyotrophic Lateral Sclerosis (ALS)

**Sponsor:** 

Mitsubishi Tanabe Pharma Development America, Inc.

525 Washington Boulevard, Suite 400

Jersey City, New Jersey 07310

**Protocol Version:** 

3.0

Protocol Date:

29 July 2022

**Original Protocol** 

Version 1.0:

02 September 2021

Amendment 1

Version 2.0:

14 December 2021

**Strictly Confidential Information** 

Mitsubishi Tanabe Pharma Corporation, Mitsubishi Tanabe Pharma Development America, Inc., their successors, and/or assignees are collectively referred to as Mitsubishi. The information contained in this protocol is the property of Mitsubishi. This information is confidential and is to be used only in connection with matters authorized by Mitsubishi and no part of it is to be disclosed to others without prior written permission from Mitsubishi.

# 1 PROTOCOL SYNOPSIS

| Name of Company Mitsubishi Tanabe P Corporation Name of Finished Pr Edaravone (MT-1186) Name of Active Ingree Edaravone (MT-1186) (3-methyl-1-phenyl-2- | oduct<br>edient | Individual Study Table Referring to Module 5 of the CTD Volume: Page: | (For National Authority Use Only) |
|---|---|---|---|
| Study Protocol Title of Study | MT-1186-A04 A Phase 3b, Multicenter, Randomized, Double-blind Extension Study to Evaluate the Continued Efficacy and Safety of Oral Edaravone Administered for an Additional Period of up to 48 Weeks Following Study MT-1186-A02 in Subjects with Amyotrophic Lateral Sclerosis (ALS) | | |
| Study Centers Study Period | Multicenter study Estimated date first subject enrolled: January 2022 Estimated date last subject completed: TBD | | |
| Phase<br>Objectives | Primary Objective: To evaluate and compare the efficacy of the following | | |
| | <ul> <li>2 dosing regimens of oral edaravone in subjects with amyotrophic lateral sclerosis (ALS), based on the time from the randomization date in Study MT-1186-A02 to at least a 12-point decrease in Revised ALS Functional Rating Score (ALSFRS-R) or death, whichever happens first, over the course of the study or until oral edaravone is commercially available in that country:</li> <li>Oral edaravone 105 mg administered once daily</li> <li>Oral edaravone 105 mg administered for 10 days followed by placebo for 18 days (regimen denoted as</li> </ul> | | |
| | on/off). Secondary Objective: • To evaluate the safety and tolerability of oral edaravone at a dose of 105 mg once daily compared to oral edaravone at a dose of 105 mg including placebo (regimen denoted as on/off) in subjects with ALS over the course of the study or | | |

| Name of Company Mitsubishi Tanabe P Corporation | harma | Individual Study Table Referring to Module 5 of the CTD | (For National Authority Use Only) |
|---|---|---|---|
| Name of Finished Pro | <u>oduct</u> | CID | |
| Edaravone (MT-1186) | | Volume: | |
| Name of Active Ingre | edient | | |
| Edaravone (MT-1186) (3-methyl-1-phenyl-2- | | Page: | |
| | until oral e country. | daravone is commer | cially available in that |
| Methodology | This is a Phase 3b, multicenter, double-blind, parallel group, randomized extension study that will evaluate the efficacy and safety of 2 treatment regimens of edaravone for an additional period of up to 48 weeks following Study MT-1186-A02 in subjects with ALS as follows: Group 1: Oral edaravone 105 mg dose once daily in each 28-day cycle for up to 48 weeks or until the drug is commercially available in that country. Group 2: Oral edaravone 105 mg dose for 10 days followed by 18-day placebo (regimen denoted as on/off) in each 28-day cycle | | evaluate the efficacy and ravone for an additional Study MT-1186-A02 in once daily in each 28-day the drug is commercially for 10 days followed by off) in each 28-day cycle |
| | 18-day placebo (regimen denoted as on/off) in each 28-day cylor up to 48 weeks or until the drug is commercially available that country. Subjects who meet Study MT-1186-A04 eligibility criteria we continue in the same treatment group/regimen that they were during Study MT-1186-A02. The Week 48 study procedures from Study MT-1186-A02 will used as the screening/entry criteria for Study MT-1186-A0 followed by a treatment period of up to an additional 48 weeks until oral edaravone is commercially available in each count whichever time period is shorter, and a safety follow-up period 2 weeks. During the conduct of Study MT-1186-A04, the dose edaravone may be adjusted or the study may be stopped based the interim futility or final analyses performed for Stu MT-1186-A02, taking into consideration the benefit and rebalance. However, unless any significant safety issue is for based on these 2 analyses, the same regimen will be kept when the study may be stopped based on these 2 analyses, the same regimen will be kept when the study may be stopped based on these 2 analyses, the same regimen will be kept when the study may be stopped based. | | old eligibility criteria will egimen that they were in addy MT-1186-A02 will be for Study MT-1186-A04, an additional 48 weeks or available in each country, safety follow-up period of may be stopped based on as performed for Study ion the benefit and risk ant safety issue is found |

| Name of Company Mitsubishi Tanabe Pharma Corporation | Individual Study Table Referring to Module 5 of the CTD | (For National<br>Authority Use Only) |
|---|---|---|
| Name of Finished Product Edaravone (MT-1186) | Volume: | |
| Name of Active Ingredient Edaravone (MT-1186) (3-methyl-1-phenyl-2-pyrazolin-5-one) | Page: | |

all personnel directly involved with the conduct of the study.

Concomitant use of riluzole is permitted throughout the course of the study when the dose and regimen remain unchanged from the screening visit evaluation of ALSFRS-R of Study MT-1186-A02 through the end-of-treatment (EOT) or early termination (ET) of Study MT-1186-A04. Dose reduction, dose interruption, or discontinuation due to the onset of adverse events (AEs), progression of dysphagia, or gastrostomy while on oral edaravone 105 mg are allowed. The use of AMX0035 will be allowed for patients in the event that it becomes commercially available via prescription in their respective country. AMX0035 should be taken at least 1 hour after MT-1186/oral edaravone dosing.

EOT assessments will occur at Week 48 (Visit 5).

For subjects who complete the double-blind treatment period, a safety follow-up telephone visit will occur at Week 50 (Visit 6).

Subjects will be allowed to change from oral administration to percutaneous endoscopic gastrostomy (PEG)/radiologically inserted gastrostomy (RIG) tube administration during the study.

Subjects who discontinue early from the study will complete the procedures listed at Week 48 (refer to Table 1 for further information) within 7 days of discontinuation. Site staff should also follow up via phone call at all remaining visits to complete the assessment for time to tracheostomy or permanent assisted mechanical ventilation, or death.

Further details can be found in the Study Schema (Figure 1).

| Name of Company Mitsubishi Tanabe Pl Corporation Name of Finished Pre Edaravone (MT-1186) | <u>oduct</u> | Individual Study Table Referring to Module 5 of the CTD Volume: | (For National Authority Use Only) |
|---|---|---|---|
| Name of Active Ingree<br>Edaravone (MT-1186)<br>(3-methyl-1-phenyl-2- | | Page: | |
| Planned Number of<br>Subjects | Approximately 300 subjects (150 subjects per dosing have successfully completed Study MT-1186-A02 through Week 48 [Visit 15]) and who meet Study M eligibility criteria will be enrolled. | | T-1186-A02 (completion |
| Diagnosis and Main Inclusion Criteria and Exclusion Criteria | 1. Subjects or provide a sparticipate in 2. Subjects musunderstand the participation 3. Subjects musurotocol rest. 4. Subjects who me from the study: 1. Subjects of acceptable 1/screening medication. agree to use Appendix 3 to 2. Subjects who pregnant (a to 1/screening to 1/ | their legally authoricing and and dated information the study. It be able (in the judgment and the study are nature of the study are nature of the study are nature and requirement at have successfully 2 visits and have been as a successfully 2 visits and have been and the following are the study are the study are the study. It is a successfully 2 visits and have been and the following are the study are sex contraception during the study are female, of chippositive pregnancy test visit. | zed representative must formed consent form to the investigator) to and all risks involved with rate and comply with all all st. y completed all Study en compliant with study g criteria will be excluded all unwilling to use an eption from the Day ther the last dose of study ually active who do not the study period. Refer to |

| Name of Company Mitsubishi Tanabe Pl Corporation Name of Finished Pro Edaravone (MT-1186) | oduct | Individual Study Table Referring to Module 5 of the CTD Volume: | (For National Authority Use Only) |
|---|---|---|---|
| Name of Active Ingree<br>Edaravone (MT-1186)<br>(3-methyl-1-phenyl-2- | | Page: | |
| | any suicidal behavior or suicidal ideation of type 4 (active suicidal ideation with some intent to act, without a specific plan) or type 5 (active suicidal ideation with specific plan and intent) based on the Columbia-Suicide Severity Rating Scale (C-SSRS) at Week 48 of Study MT-1186-A02. 4. Subjects who are not eligible to continue in the study, as judged by the Investigator in conjunction with the MTDA medical monitor. 5. Subjects who are unable to take their medications orally or through a PEG/RIG tube. | | to act, without a specific eation with specific plan -Suicide Severity Rating y MT-1186-A02. continue in the study, as unction with the MTDA |
| Endpoints | Primary Efficacy Endpoint: | | |
| | <ul> <li>Time from the randomization date in Study MT-1186-A02 t at least a 12-point decrease in ALSFRS-R or death whichever happens first.</li> <li>Secondary Efficacy Endpoints:</li> <li>The Combined Assessment of Function and Surviva (CAFS) score at all visits from baseline in Stud MT-1186-A02 to the end of Study MT-1186-A04</li> </ul> | | ALSFRS-R or death, Function and Survival om baseline in Study MT-1186-A04 |
| | • Change in the Amyotrophic Lateral Sclerosis Assessment Questionnaire 40 score at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04 | | s from baseline in Study |
| | • Change in ALSFRS-R score at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04 | | |
| | • Time from the randomization date in Study MT-1186-A02 to death, tracheostomy, or permanent assisted mechanical ventilation (≥23 hours/day) | | |
| | • Time from the randomization date in Study MT-1186-A02 death or permanent assisted mechanical ventilation (≥23 hours/day) | | |
| | • Time from the death | he randomization date | in Study MT-1186-A02 to |

| Name of Company Mitsubishi Tanabe Pharma Corporation | | Individual Study Table Referring to Module 5 of the CTD | (For National Authority Use Only) |
|---|---|---|---|
| Name of Finished Pr | <u>oduct</u> | CID | |
| Edaravone (MT-1186) | ) | Volume: | |
| Name of Active Ingre | <u>edient</u> | | |
| Edaravone (MT-1186)<br>(3-methyl-1-phenyl-2- | | Page: | |
| | Exploratory Effi | cacy Endpoints: | |
| | | Study MT-1186-A02 | (SVC) at all visits from to the end of Study |
| | | ody weight at all visit<br>2 to the end of Study N | s from baseline in Study<br>//T-1186-A04 |
| | • King's ALS Clinical Stage derived from ALSFRS-R score and death at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04 | | |
| | Safety Endpoints: The following endpoints will be assessed for safety: | | |
| · | AEs, adverse drug reactions, and treatment-emergent adverse events (TEAEs; e.g., grade, incidence, severity) | | |
| | Physical examination | | |
| | • 12-lead electrocardiogram (ECG) parameters | | |
| · | • Vital signs (heart rate, respiratory rate, sitting systolic and diastolic blood pressure, and axillary, oral, temporal [skin-based], or tympanic body temperature) | | |
| | • Laboratory safety assessments (e.g., hematology, chemistry, and urinalysis) | | |
| | • C-SSRS | | |
| Statistical Methods | The analysis undertaken for Study MT-1186-A04 will include data from the beginning (baseline) of Study MT-1186-A02 until the end of Study MT-1186-A04. The data will also include information for subjects who early terminated during Study MT-1186-A02 or decided not to continue into Study MT-1186-A04. | | |

| Name of Company Mitsubishi Tanabe Pharma Corporation | Individual Study Table Referring to Module 5 of the CTD | (For National Authority Use Only) |
|---|---|---|
| Name of Finished Product Edaravone (MT-1186) | Volume: | |
| Name of Active Ingredient Edaravone (MT-1186) (3-methyl-1-phenyl-2-pyrazolin-5-one) | Page: | |

# **Primary Estimand**

The primary estimand construction elements are:

- Treatment of interest: The initially randomized treatment Group 1 (edaravone daily) to be compared with Group 2 (edaravone on/off) for up to 96 weeks.
- Population: Subjects with ALS as defined in the analysis set.
- Variable: Time from the randomization date in Study MT-1186-A02 to at least a 12-point decrease in ALSFRS-R or death, whichever happens first.
- Inter-current event (ICE) handling strategy
  - ➤ ICE1 Additional AMX0035 treatment up to 96 weeks double-blind treatment period will be handled using treatment policy strategy.
  - ➤ ICE2 Death will be handled within the primary endpoint derivation using Composite variable strategy.
- Population-level summary: the Kaplan-Meier estimates and the hazard ratio between Group 1 and Group 2 will be derived from the Kaplan-Meier plot and Cox PH regression, respectively.

The treatment effect on the primary endpoint taking death event (ICE2) into account is attributed regardless of the use of additional AMX0035 treatment (ICE1).

# **Secondary Estimand**

The secondary estimand will be tested as supportive analysis for the primary endpoint.

The secondary estimand construction elements are:

- Treatment of interest: as specified for the primary estimand.
- Population: as specified for the primary estimand.

| Name of Company Mitsubishi Tanabe Pharma Corporation | Individual Study Table Referring to Module 5 of the | (For National Authority Use Only) |
|---|---|---|
| Name of Finished Product Edaravone (MT-1186) | CTD Volume: | |
| Name of Active Ingredient Edaravone (MT-1186) (3-methyl-1-phenyl-2-pyrazolin-5-one) | Page: | |

- Variable: as specified for the primary estimand.
- ICE handling strategy
  - ➤ ICE1 Additional AMX0035 treatment up to 96 weeks double-blind treatment period will be handled using hypothetical strategy.
  - ➤ ICE2 Death will be handled within the primary endpoint derivation using composite variable strategy.
- Population-level summary: as specified for the primary estimand.

The above estimand will also be tested when the primary endpoint event is censored if it occurs after ICE1 (Additional AMX0035 treatment). In this estimand, the treatment effect will be attributed as if AMX0035 treatment had not been available.

### **Determination of Sample Size:**

The sample size for this study is not based on a formal statistical calculation. In total, approximately 300 subjects who have successfully completed Study MT-1186-A02 will be enrolled in this study. However, data from 380 subjects (190 subjects per group) randomized in Study MT-1186-A02 will be included for all analyses. Using Study MT-1186-A02 and MT-1186-A04 survival data, the planned sample size of 190 subjects per group initially randomized in Study MT-1186-A02 will have 70% power to detect a statistically significant result if the true hazard ratio between edaravone 105 mg daily (test) and edaravone 105 mg on/off regimen (control) in the primary endpoint is 0.775, which means 22.5% risk reduction in the hazard due to daily treatment, assuming 65% survival rate at Week 48 for the control group. This calculation of 70% power assumes a 2-sided alpha of 20% based on a rare disease condition (Hilgers RD et al., 2016), using the log-rank test and a follow-up time of up to 48 weeks in Study MT-1186-A04.

| Name of Company Mitsubishi Tanabe Pharma Corporation | Individual Study Table Referring to Module 5 of the CTD | (For National<br>Authority Use Only) |
|---|---|---|
| Name of Finished Product Edaravone (MT-1186) | Volume: | |
| Name of Active Ingredient Edaravone (MT-1186) (3-methyl-1-phenyl-2-pyrazolin-5-one) | Page: | |

### **Baseline Definition:**

The data collected before the first study drug dose administration date in Study MT-1186-A02 will be used as the baseline for statistical analysis in Study MT-1186-A04.

# **Analysis Sets**

The statistical analysis will be based on separate analysis sets, defined as follows:

### Randomized Set

The randomized set is defined as all of the subjects randomized in Study MT-1186-A02. The subjects will be grouped by the planned treatment allocation (as randomized).

# **Efficacy Analysis Set**

The full analysis set (FAS) is defined as all of the subjects randomized in Study MT-1186-A02, who received at least 1 dose of study medication in Study MT-1186-A02 and had any efficacy data collected after randomization. Subjects in the FAS will be grouped and analyzed based on the planned treatment allocated (as randomized). Efficacy endpoints will be analyzed using the FAS.

# Safety Analysis Set

The Safety Analyses Set (SAF) is defined as all of the subjects randomized in Study MT-1186-A02, and who received at least 1 dose of study drug in Study MT-1186-A02. Subjects will be grouped and analyzed based on the actual treatment received. Safety endpoints will be analyzed using the SAF by treatment group.

### Statistical Methods

In general, continuous variables will be summarized descriptively using the number of observations (n), mean, standard deviation, median, minimum, and maximum.

| Name of Company Mitsubishi Tanabe Pharma Corporation | Individual Study Table Referring to Module 5 of the CTD | (For National Authority Use Only) |
|---|---|---|
| Name of Finished Product Edaravone (MT-1186) | Volume: | |
| Name of Active Ingredient Edaravone (MT-1186) (3-methyl-1-phenyl-2-pyrazolin-5-one) | Page: | |

Categorical variables will be summarized using frequency counts and percentages.

# Type I Error

Since no formal hypothesis was formulated, type I error will not be controlled. Unless otherwise specified, all statistical tests for the primary endpoint and the other endpoints will be done as 2-sided with a nominal 20% and 5% significance level, respectively. Point estimates of treatment differences will be accompanied with 2-sided 80% and 95% confidence intervals (CIs) where applicable, respectively.

# **Study Medication Exposure**

The duration of exposure in days will be calculated as follows:

Date of last dose of edaravone in Study MT-1186-A04 – date of first dose of edaravone in Study MT-1186-A02 + 1

If the date of first dose or the date of last dose cannot be determined, the duration calculation will not be completed. The duration of exposure will be summarized using descriptive statistics.

All exposure data will be listed. Interruptions and compliance are not considered for the duration of exposure.

# Primary Analysis for the Primary Efficacy Endpoint

Data of time from randomization in Study MT-1186-A02 to at least a 12-point decrease in ALSFRS-R or death will be included regardless of AMX0035 use (ICE1). In other words, data following AMX0035 treatment will be used in the analysis and will not be censored.

The primary efficacy endpoint associated with the study estimand will be analyzed on the randomized set using Kaplan-Meier estimates, 2-sided alpha with a nominal 20% significance level and 80% CIs. The comparison between

| Name of Company Mitsubishi Tanabe Pharma Corporation | Individual Study Table Referring to Module 5 of the | (For National Authority Use Only) |
|---|---|---|
| Name of Finished Product Edaravone (MT-1186) | CTD Volume: | |
| Name of Active Ingredient Edaravone (MT-1186) (3-methyl-1-phenyl-2-pyrazolin-5-one) | Page: | |

Treatment Group 2 versus Treatment Group 1 will be performed using a log rank test with MT-1186-A02 randomization strata of ALSFRS-R rate of decline score from the MT-1186-A02 screening period (2 levels strata of -1,-2 or -3,-4) and the geographical region (3 levels strata of Europe, America, or Asia Pacific). Subjects without events during treatment will be right censored at the date of last study visit.

# Supportive Analyses for the Primary Endpoint

The primary efficacy endpoint will also be analyzed using the Cox Proportional Hazard (COX PH) Model with terms for treatment as explanatory variable and baseline ALSFRS-R score, and the MT-1186-A02 randomization strata as covariates.

This statistical test will be done as 2-sided with a nominal 20% significance level. Point estimates of treatment differences will be accompanied with 2-sided 80% CIs.

# Supportive Analysis for the Secondary Estimand

The primary analysis will be repeated when the event of interest is censored if it occurred after initiation of AMX0035 treatment, using the Inverse Probability of Censoring Weighting (IPCW by Robins JM, Finkelstein et all, 2000) to adjust for non-random time-dependent covariates.

### **Efficacy Analyses for Secondary Endpoints**

CAFS analysis ranks clinical outcomes on the basis of survival time and change in the ALSFRS-R score will be analyzed at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04. In this analysis, a subject's score will be calculated by comparing each subject to every other subject within each treatment group in the study, resulting in a score of +1 if the outcome was better than the subject being compared, -1 if worse, and 0 if the same. The subject's score will then be calculated by summing up their comparison to all of the other subjects within each treatment group in the study as CAFS score.

| Name of Company Mitsubishi Tanabe Pharma Corporation | Individual Study Table Referring to Module 5 of the CTD | (For National Authority Use Only) |
|---|---|---|
| Name of Finished Product Edaravone (MT-1186) | Volume: | |
| Name of Active Ingredient Edaravone (MT-1186) (3-methyl-1-phenyl-2-pyrazolin-5-one) | Page: | |

A subject who dies earlier than the comparator subject will be given a comparison score of -1. For a subject who discontinues early for a reason other than death, that subject and the comparator's score will be based on the change from baseline of the ALSFRS-R score at the latest timepoint at which they both have an ALSFRS-R score. In general, these comparisons will result in subjects who die being assigned the worst scores and ranked according to the time of death. Subjects who survive and complete the study will be ranked more favorably than subjects who die. The CAFS score at all visits will be evaluated at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04 using an analysis of covariance model with treatment group and Study MT-1186-A02 randomization strata as fixed effects, and baseline ALSFRS-R total score as covariate. The difference between the 2 treatment groups in the CAFS scores will be also compared using the generalized Gehan-Wilcoxon test as a sensitivity analysis.

The following sequence of parametric and semi-parametric models will be conducted to estimate the clinical benefit:

- Mixed-effect model for repeated measure (MMRM) as specified below.
- COX PH model as specified above.

Change in ALSFRS-R score will be analyzed at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04 using MMRM with terms for baseline ALSFRS-R score, Study MT-1186-A02 randomization strata, treatment, visit, and treatment-by-visit interaction. The unstructured covariance matrix will be used to model the within-subject errors. Denominator degrees of freedom will be estimated using Kenward-Roger's approximation. The least-squares mean estimates for the mean change from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04, as well as the difference of the estimates between oral edaravone 105 mg daily

| Name of Company Mitsubishi Tanabe Pharma Corporation | Individual Study Table Referring to Module 5 of the CTD | (For National<br>Authority Use Only) |
|---|---|---|
| Name of Finished Product Edaravone (MT-1186) | Volume: | |
| Name of Active Ingredient Edaravone (MT-1186) (3-methyl-1-phenyl-2-pyrazolin-5-one) | Page: | |

versus oral edaravone 105 mg on/off regimen, will be displayed with their corresponding standard errors, p-values, and 95% CI.

# Efficacy Analyses for Other Secondary Exploratory Endpoints

The following endpoints with continuous values will be analyzed using the same method (MMRM) and the same survival analysis as specified above:

- 1. Time from the randomization date in Study MT-1186-A02 to death, tracheostomy, or permanent assisted mechanical ventilation (≥23 hours/day)
- 2. Change in %SVC at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04
- 3. Change in body weight from at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04
- 4. Time from the randomization date in Study MT-1186-A02 to death or permanent assisted mechanical ventilation (≥23 hours/day)
- 5. Time from the randomization date in Study MT-1186-A02 to death
- 6. Change in ALSAQ40 at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04

# **Efficacy Analyses for Other Exploratory Endpoints**

King's ALS Clinical Stage will be derived from ALSFRS-R score and death. The frequency and percent for King's ALS Clinical Stage at each visit will be provided by each treatment group using shift tables.

# Safety Endpoints and Analyses

An AE will be considered a TEAE if:

| Name of Company Mitsubishi Tanabe Pharma Corporation | Individual Study Table Referring to Module 5 of the CTD | (For National Authority Use Only) |
|---|---|---|
| Name of Finished Product Edaravone (MT-1186) | Volume: | |
| Name of Active Ingredient Edaravone (MT-1186) (3-methyl-1-phenyl-2-pyrazolin-5-one) | Page: | |

- 1) The AE was not present before the first dose in Study MT-1186-A02 but started after administration of the first dose of study drug in Study MT-1186-A02, or
- 2) The AE was present before the first dose in Study MT-1186-A02 but increased in severity following administration of the first dose of study drug in Study MT-1186-A02.

TEAEs will be coded using the latest available version of the Medical Dictionary for Regulatory Activities (MedDRA) and will be summarized in incidence tables by System Organ Class (SOC) and Preferred Term (PT). The numbers and proportions of subjects with TEAEs will be calculated for each treatment group by SOC and PT.

The following summaries will be presented:

- TEAEs by SOC and PT
- TEAEs by SOC, PT, and severity
- TEAEs by SOC, PT, and drug relationship
- TEAEs leading to discontinuation of study drug by SOC and PT
- TEAEs leading to death by SOC and PT
- TEAEs related to study drug by SOC, PT, and severity
- TEAEs of Peripheral Neuropathy Standardized MedDRA query by SOC and PT
- Serious TEAEs by SOC and PT
- Serious TEAEs related to study drug by SOC and PT

For each of the summaries, multiple occurrences of the same event within a subject will be counted once in the summaries by SOC and PT; multiple occurrences of the same event within a subject will be counted once in the maximum severity category (severe>moderate>mild) and/or maximum study drug relationship category (reasonable possibility/no reasonable

| Name of Company Mitsubishi Tanabe P Corporation | harma | Individual Study Table Referring to Module 5 of the CTD | (For National Authority Use Only) |
|---|---|---|---|
| Name of Finished Pr | <u>oduct</u> | <u> </u> | |
| Edaravone (MT-1186) | | Volume: | |
| Name of Active Ingre<br>Edaravone (MT-1186)<br>(3-methyl-1-phenyl-2- | | Page: | |
| | , | • | found to be missing, the uted for that particular |
| | | or listed according to | tions will be summarized the data type and will |
| | <ul><li>12-lead ECG</li><li>Vital signs</li><li>Clinical labora</li><li>C-SSRS</li></ul> | atory assessments | |



Abbreviation: EOS = end-of-study; EOT = end-of-treatment; ET = early termination.

- Subjects will receive oral edaravone at a dose of 105 mg administered once daily in each 28 Day Cycle or a dose of 105 mg administered for 10 days, followed by placebo for 18 days in each 28 Day Cycle. The dose of edaravone should be taken following an overnight fast and at least 1 to 2 hours before the morning meal. Day 1 is equal to the Week 48 visit of Study MT-1186-A02. æ.
  - .

# Figure 1: Study Schema

Page 17 of 89

Schedule of Assessments Table 1:

| Assessment | | | | | | |
|---|---|---|---|---|---|---|
| Week (window) | Day 1 | 12 | 24 | 36 | 48 | 20 |
| | (Based on Week 48 | (± 7D) | (± 7D) | (± 7D) | (± 7D) | (± 7D) Telephone Visit |
| | procedures from<br>Study MT-1186-A02) | Telephone Visit | | Telephone Visit | EOT/ET <sup>a</sup> | EOS |
| Cycle | 1 | 4 | 7 | 10 | | |
| Visit | 1 | 2 | 3 | 4 | છ | 9 |
| Informed consent | X | | | | | |
| Eligibility criteria | X | | | | | |
| Demographics <sup>b</sup> | X | | | | | |
| Vital signs <sup>c</sup> | X | | X | | × | |
| Full Physical examination <sup>d</sup> | X | | | | × | |
| Routine physical examination <sup>d</sup> | | | × | | | |
| 12-lead ECG <sup>e</sup> | X | | X | | × | |
| Body weight | X | | × | | X | |
| Time to event of death, tracheostomy or permanent assisted mechanical ventilation <sup>f</sup> | X | × | × | × | × | × |
| Hematology <sup>g</sup> | X | | X | | × | |
| Chemistry <sup>h</sup> | X | | × | | × | |
| Urinalysis <sup>i</sup> | X | | × | | × | |
| Serum Pregnancy Test (WOCP only) | X | | × | | × | |
| Urine Pregnancy Test (WOCP only) $^{\rm j}$ | X | | | | | |
| Dispense edaravone k | X | | X | | | |
| ALSFRS-R | X | × | × | × | × | |
| ALSAQ40 | X | | × | | × | |
| Slow Vital Capacity | X | | × | | × | |
| C-SSRS | X | | × | | × | |
| Adverse events | X | X | × | × | × | × |

Version 3.0, 29 July 2022

Confidential

Page 18 of 89

| Assessment | | | | | | |
|---|---|---|---|---|---|---|
| Week (window) | Day 1 (Bosed on Wools 48 | 12 | | 36 | 48<br>£ | 50<br>(+ 7D) Talenhone Vicit |
| | procedures from Study MT-1186-A02) | (± /D)<br>Telephone Visit | (T/ ±) | (= /D)<br>Telephone Visit | EOT/ET <sup>a</sup> | EOS |
| Cycle | 1 | 4 | 7 | 10 | | |
| Visit | 1 | 2 | 3 | 4 | 5 | 9 |
| Concomitant medications | X | X | X | X | X | X |
| Medication Compliance Assessment <sup>1</sup> | X | X | X | X | × | |

Abbreviation: AE = adverse event; ALSAQ = Amyotrophic Lateral Sclerosis Assessment Questionnaire; ALSFRS-R = Revised Amyotrophic Lateral Sclerosis Functional Rating Scale; C-SSRS = Columbia-Suicide Severity Rating Scale; D = Day; ECG = Electrocardiogram; EOS = End-of-study; EOT = End-of-treatment; ET = Early Termination; WOCP = women of childbearing potential.

- Subjects who withdraw from the study will complete the procedures listed in ET within 7 days of study discontinuation. ä
  - Demographics will include age, sex, race, and ethnicity. <u>ن</u>
- Vital signs will include sitting systolic and diastolic blood pressure, heart rate, respiratory rate, and axillary, oral, temporal (skin-based), or tympanic body temperature. ပ
- 1. A full physical examination will consist of an assessment of the major body parts and systems: abdominal, cardiovascular, general appearance, head, eyes, ears/nose/throat, lymph nodes, musculoskeletal, neck, neurological, dermatological, respiratory, and other.
  - Routine physical examination will include abdominal, cardiovascular, general appearance, respiratory, neurological, and other.
- A 12-lead ECG will be performed after the subject has rested for at least 5 minutes in a supine position. The ECG must include the following measurements: R wave to Investigator will perform an overall evaluation of the ECG for safety purposes and the recording will be reported as 'normal', 'abnormal clinically significant (CS)', or R wave (RR) interval, heart rate, QRS, and QT. If available, corrected QT interval by Bazett, and corrected QT interval by Fridericia should also be recorded. The 'abnormal not clinically significant (NCS)'. Abnormalities of clinical significance will be reported as AEs.
  - Events are time to death, tracheostomy, or permanent assisted mechanical ventilation ( $\geq 23$  hours/day). If a subject discontinues early from the study, study sites must follow-up with phone calls at all remaining visits.
    - To include: red blood cell count, hemoglobin, hematocrit value, white blood cell count with differential, and platelet count.
- c-reactive protein, creatine kinase, total cholesterol, triglycerides, blood urea nitrogen, bicarbonate, serum glucose, serum creatinine level, uric acid, sodium, potassium, To include: albumin, total protein, aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase, alkaline phosphatase, total bilirubin, direct bilirubin, chloride, calcium, cystatin-C, and vitamin B6. <u>ئە</u> بىز
  - To include protein, glucose, occult blood, urobilinogen, white blood cells, and bilirubin.
- For female subjects of childbearing potential (WOCP) only, urine beta-human chorionic gonadotropin test will be conducted.
- placebo for 18 days (regimen denoted as on/off) in Cycles 1 through 12, following an overnight fast, and subjects must continue to fast at least 1 to 2 hours post-dose Subjects will receive oral edaravone 105 mg once daily in each 28 Day Cycle (Cycles 1 through 12) or oral edaravone 105 mg administered for 10 days followed by before the next meal (e.g., breakfast)
- Screening/Day 1 drug compliance should be assessed as part of Study MT-1186-A02/Week 48 visit. Once a subject is eligible to enroll in Study MT-1186-A04, drug compliance should be assessed on a per cycle basis by site staff via study phone calls (Weeks 12 and 36) or during the in-clinic visits.

| 2 TABLE OF CONTENTS | |
|---|---|
| 1 PROTOCOL SYNOPSIS | 2 |
| TABLE OF CONTENTS | |
| 3 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 24 |
| 4 SIGNATURES | |
| 5 SPONSOR AND ADMINISTRATIVE STRUCTURE | |
| 6 INTRODUCTION | |
| 6.1 Background | |
| 6.1.1 Known Potential Benefits and Previous Experience with the Oral Formulation | |
| 6.1.1.1 Benefits of Edaravone | 32 |
| 7 STUDY OBJECTIVES, ENDPOINTS, and HYPOTHESES | 36 |
| 7.1 Study Objectives | 36 |
| 7.1.1 Primary Objective | |
| 7.1.2 Secondary Objective | |
| 7.2 Study Endpoints | 37 |
| 7.2.1 Primary Efficacy Endpoint | 37 |
| 7.2.2 Secondary Efficacy Endpoints | 37 |
| 7.2.3 Exploratory Efficacy Endpoints | 37 |
| 7.2.4 Safety Endpoints | 37 |
| 7.2.5 Hypothesis | |
| 8 STUDY DESIGN | |
| 8.1 Overall Study Design | 38 |
| 8.2 Rationale for Study Design | 39 |
| 8.2.1 Risk/Benefit Assessment | |
| 8.2.2 Rationale for Dose Selection | |
| 8.2.3 Independent Data Monitoring Committee | |
| · | 41<br>11 |
| 9.2 Recruitment Methods | |
| 9.4 Exclusion Criteria | |
| 9.5 Screen Failures | |
| 9.6 Withdrawal of Individual Subjects | |
| 10 STUDY PLAN | 44 |
| 10.1 Description of Study Periods | 44 |
| 10.1.1 Double-blind Treatment Period. | |
| 10.1.2 Optional Open Label Treatment Period | |
| 10.1.3 End-of-Treatment/Early Termination Period | 44 |
| 10.1.4 Safety Follow-up Period | 45 |
| 10.1.5 End-of-Study Options | 45 |
| 10.1.6 Unscheduled Visits | 45 |
| 11 STUDY PROCEDURES | |
| 11.1 Concomitant Medications | |
| 11.2 Prohibited Concomitant Medications | |
| 11.3 Permitted Concomitant Medications | 46 |

| 12 EFFICACY ASSESSMENTS | 47 |
|---|---|
| 12.1 Primary Efficacy Assessment | 47 |
| 12.1.1 ALS Functional Rating Scale | 47 |
| 12.2 Secondary Efficacy Assessment | 47 |
| 12.2.1 Combined Assessment of Function and Survival Score | 47 |
| 12.2.2 Time to Death, Tracheostomy, or Permanent Assisted Ventilation | 47 |
| 12.3 Exploratory Efficacy Assessment | |
| 12.3.1 Slow Vital Capacity | |
| 12.3.2 Body Weight | 48 |
| 12.3.3 King's ALS Clinical Stage Derived from ALSFRS-R Score and Death Event | |
| 13 SAFETY ASSESSMENTS | |
| 13.1 Physical Examination | |
| 13.2 Vital Signs | |
| 13.3 Body Weight | |
| 13.4 12-lead Electrocardiogram | |
| 13.5 Clinical Laboratory Tests | |
| 13.5.1 Hematology | |
| 13.5.2 Blood Chemistry | |
| 13.5.3 Urinalysis (Qualitative) | |
| 13.5.4 Pregnancy Test | |
| 13.6 Columbia-Suicide Severity Rating Scale (C-SSRS) | |
| 14 STUDY DRUG TREATMENT | |
| 14.1 Investigational Medicinal Product | |
| 14.1.1 Drug Product | |
| 14.1.2 Study Drug Supply | |
| 14.1.3 Formulation, Packaging, and Labeling | |
| 14.1.4 Shipping, Receipt, Handling, and Storage | |
| 14.1.5 Dispensing | 52 |
| 14.1.6 Study Medication Accountability | 52 |
| 14.1.7 Disposal and Destruction | 52 |
| 14.2 Dosing of Edaravone or Placebo | |
| 14.3 Treatment Compliance | |
| 14.4 Subject Identification | |
| 14.5 Procedures for Assigning Subjects to Treatment Groups | |
| 14.6 Maintenance of the Study Blind and Unblinding | |
| 14.7 Dose Adjustment Criteria | |
| 15 ADVERSE EVENT MANAGEMENT | |
| 15.1 Adverse Event | |
| 15.2 Serious Adverse Event | |
| 15.3 Severity of Adverse Events | |
| 15.4 Relationship of Adverse Events to Investigational Medicinal Product | 56 |
| 15.5 Clinical Laboratory Abnormalities and Other Abnormal Assessments | |
| 15.6 Recording and Reporting of Adverse Events | |
| 15.7 Recording and Reporting of Serious Adverse Events | |
| 15.8 Follow-up of Adverse Events | |
| 15.9 Pregnancy | 58 |

| 15.10 Reference Safety Information | 58 |
|---|---|
| 15.11 Overdose | |
| 16 DATA COLLECTION AND PROCESSING | |
| 16.1 Data Collection | |
| 16.2 Case Report Form | |
| 16.3 Data Processing | 61 |
| 17 STATISTICAL METHODS and PLANNED ANALYSES | |
| 17.1 Study Estimands | |
| 17.2 Determination of Sample Size | |
| 17.3 Analysis Sets | 64 |
| 17.4 Statistical Analyses | 64 |
| 17.4.1 General Considerations | |
| 17.4.2 Data Handling | 64 |
| 17.4.2.1 Definition of Baseline for the Efficacy and Safety Endpoints | 64 |
| 17.4.2.2 Handling of Time Point Data in Analyses Performed by Measurement Time | |
| Point (Analysis Visit Windows) | 64 |
| 17.4.2.3 Handling of Reference Values and Indeterminate Values for Clinical Laboratory | |
| Test Parameters | |
| 17.4.3 Statistical Analysis Method | |
| 17.4.3.1 Subject Disposition | 65 |
| 17.4.3.2 Concomitant Medications | |
| 17.4.4 Study Medication Exposure | 65 |
| 17.4.5 Efficacy Analysis | 66 |
| 17.4.5.1 Primary Efficacy Analysis | 66 |
| 17.4.5.2 Supportive Analyses for the Primary Efficacy Endpoint | 66 |
| 17.4.5.3 Supportive Analysis for the Secondary Estimand | 66 |
| 17.4.5.4 Efficacy Analyses for Secondary Endpoints | 66 |
| 17.4.5.5 Efficacy Analyses for Other Secondary Exploratory Endpoints | |
| 17.4.5.6 Efficacy Analyses for Other Exploratory Endpoints | |
| 17.4.5.7 Type I Error Control | 68 |
| 17.4.5.8 Safety Analyses | 68 |
| 17.4.5.9 Other Safety Analyses | 69 |
| 18 STUDY MANAGEMENT AND ETHICAL AND REGULATORY REQUIREMENT | |
| 18.1 Good Clinical Practice | |
| 18.2 Investigator Responsibilities | 70 |
| 18.2.1 Informed Consent Form | |
| 18.2.2 Ethical and Regulatory Approval | 71 |
| 18.2.3 Source Document Requirements and Document Access During the Study | 72 |
| 18.2.4 Study Records Retention | 72 |
| 18.3 Study Monitoring | 72 |
| 18.4 Quality Assurance and Auditing | |
| 18.5 End-of-study and Site Closure | 73 |
| 18.6 Premature Discontinuation of the Study | |
| 18.7 Liability and Insurance | |
| 19 DISCLOSURE OF DATA | |
| 19.1 Confidentiality | /5 |

# Protocol MT-1186- A04

| 19.2 Publicati | on | 75 |
|---|---|---|
| | REFERENCES | |
| 21 APPENI | DICES | 78 |
| | El Escorial Revised Criteria For Diagnosis Of Amyotrophic Lateral Scleros | |
| 11 | (EXAMPLE) | |
| Appendix 2 | ALS Functional Rating Scale- Revised (ALSFRS-R) (EXAMPLE) | 80 |
| Appendix 3 | Subject Contraception | |
| Appendix 4 | Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ) 40 | |
| 11 | (example) | 83 |
| Appendix 5 | Columbia-Suicide Severity Rating Scale (example) | 87 |
| | LIST OF TABLES | |
| Table 1: | Schedule of Assessments | 18 |
| Table 2: | Emergency Contact Information | |
| Table 3: | Investigational Product | 53 |
| 2.00.00 | | |
| | LIST OF FIGURES | |
| Figure 1: | Study Schema | 17 |

# 3 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation or Specialist Term | Explanation |
|---|---|
| AE | Adverse Event |
| AIS | Acute Ischemic Stroke |
| ALS | Amyotrophic Lateral Sclerosis |
| ALSFRS-R | Revised Amyotrophic Lateral Sclerosis Functional Rating Scale |
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| ATS | American Thoracic Society |
| AUC | Area Under the Concentration-time Curve |
| AUC <sub>0-24h</sub> | Area Under the Concentration-time Curve From Time 0 to 24 Hours |
| $\mathrm{AUC}_{0	imes}$ | Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity |
| BCRP | Breast Cancer Resistance Protein |
| CAFS | Combined Assessment of Function and Survival |
| CFR | Code of Federal Regulations |
| CHMP | Committee for Medicinal Products for Human Use |
| CI | Confidence Interval |
| $C_{\max}$ | Maximum Concentration |
| COVID-19 | Coronavirus Disease 2019 |
| COX PH | Cox Proportional Hazard |
| CRO | Contract Research Organization |
| CS | Clinically Significant |
| CSR | Clinical Study Report |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| СҮР | Cytochrome P450 |
| DDI | Drug-drug Interaction |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EOS | End-of-study |
| ЕОТ | End-of-treatment |
| ERS | European Respiratory Society |

| Abbreviation or Specialist Term | Explanation |
|---|---|
| ET | Early Termination |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| ICE | Inter-current event |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IEC | Independent Ethics Committee |
| IMP | Investigational Medicinal Product |
| IRB | Institutional Review Board |
| IV | Intravenous |
| IVRS | Interactive Voice Response System |
| IWRS | Interactive Web Response System |
| LAR | Legally Authorized Representative |
| LMN | Lower Motor Neuron Degeneration |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed-effect Model for Repeated Measure |
| MTDA | Mitsubishi Tanabe Pharma Development America, Inc. |
| NCS | Not Clinically Significant |
| OAT | Organic Anion Transporter |
| PEG | Percutaneous Endoscopic Gastrostomy |
| PK | Pharmacokinetic |
| PT | Preferred Term |
| RIG | Radiologically Inserted Gastrostomy |
| RR | R Wave to R Wave |
| QTcB | Corrected QT Interval by Bazett |
| QTcF | Corrected QT Interval by Fridericia |
| SAE | Serious Adverse Event |
| SAF | Safety Analysis Set |
| SAP | Statistical Analysis Plan |
| SOC | System Organ Class |
| SUSAR | Suspected Unexpected Serious Adverse Reactions |
| SVC | Slow Vital Capacity |

# Protocol MT-1186-A04

| Abbreviation or Specialist Term | Explanation |
|---------------------------------|-------------------------------------------|
| TEAE | Treatment-emergent Adverse Event |
| t <sub>max</sub> | Time to Maximum Concentration |
| ULN | Upper Limit of Normal |
| US | United States |
| USPI | United States Prescribing Information |
| WBC | White Blood Cell |
| WMA | World Medical Association |
| WHO DD | World Health Organization Drug Dictionary |

# 4 SIGNATURES

# **SPONSOR'S RESPONSIBLE SIGNATORY**

Protocol Number: MT-1186-A04

A Phase 3b, Multicenter, Randomized, Double-blind Extension Study to Evaluate the Continued Efficacy and Safety of Oral Edaravone Administered for an Additional Period of up to 48 Weeks Following Study MT-1186-A02 in Subjects with Amyotrophic Lateral Sclerosis (ALS)

The Protocol has been designed according to the International Council for Harmonisation (ICH) Tripartite Guideline for Good Clinical Practice (GCP), the Declaration of Helsinki (Fortaleza, Brazil, 2013) and the Code of Federal Regulations (CFR). It has undergone both medical and scientific review by competent Sponsor personnel. The study will be initiated at the site(s) only after Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approval of the necessary essential documents and study procedures will not be initiated until the subject or their legally authorized representative has signed the approved Subject Information and Informed Consent Form(s) (ICF).



# **STATISTICIAN**

### Protocol Number: MT-1186-A04

A Phase 3b, Multicenter, Randomized, Double-blind Extension Study to Evaluate the Continued Efficacy and Safety of Oral Edaravone Administered for an Additional Period of up to 48 Weeks Following Study MT-1186-A02 in Subjects with Amyotrophic Lateral Sclerosis (ALS)

The Protocol has been designed according to the International Council for Harmonization (ICH) Tripartite Guideline for Good Clinical Practice (GCP) and has undergone statistical review.

### Statistician:

\*NOTE: Electronic Signature is located on the last page of the document.



# SIGNATURE PAGE (PRINCIPAL INVESTIGATOR)

Protocol Number: MT-1186-A04

A Phase 3b, Multicenter, Randomized, Double-blind Extension Study to Evaluate the Continued Efficacy and Safety of Oral Edaravone Administered for an Additional Period of up to 48 Weeks Following Study MT-1186-A02 in Subjects with Amyotrophic Lateral Sclerosis (ALS)

I confirm that I have read this Protocol and understand its contents. I agree to fully comply with its requirements. I understand it and will conduct the study in accordance with the procedures described in this protocol and the principles of GCP as described in 21 CFR, Parts, 50, 56, and 312, as well as any applicable local requirements.

I agree to make no changes to the conduct of the study as defined by the Protocol without the prior authorization of Mitsubishi Tanabe Pharma Development America, Inc. in the form of a Protocol Modification and without the appropriate Federal Drug Administration and Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approvals.

| Address of Institution: | <br> |
|-------------------------|------|
| Signed: Print Name: | |
| | <br> |
| Title: | |
| Date: | |

# 5 SPONSOR AND ADMINISTRATIVE STRUCTURE

**Table 2:** Emergency Contact Information

| Role in Study | Name | Address and Telephone<br>Number |
|---------------------------------|------|---------------------------------|
| Global Clinical Study<br>Leader | | |
| Global Medical Lead | | |
| Drug Safety Physician | | |

# 6 INTRODUCTION

# 6.1 Background

Amyotrophic lateral sclerosis (ALS) is a rare disease, which causes progressive and fatal neurodegenerative disorders.<sup>1,2,3</sup> Currently incurable, respiratory failure leads to death in a mean time of 2 to 4 years for the majority of subjects with ALS after the onset of the first symptoms. However, 5% to 10% of subjects may survive for a decade or more.<sup>4</sup>

Early stages of the disease appear in several forms and the lack of biological markers make ALS particularly difficult to diagnose. ALS is typically diagnosed by excluding other possible diseases. The El Escorial criteria have been developed and revised by the World Federation of Neurology<sup>5,6</sup>; the criteria are based on clinical signs and electrophysiological and neuroimaging evidence, and allow for the diagnosis of ALS in 5 categories: definite ALS, probable ALS, probable laboratory-supported ALS, possible ALS, or suspected ALS.

ALS is a disease of unknown cause in which primary motor neurons (upper motor neurons) and secondary motor neurons (lower motor neurons) degenerate and are lost selectively and progressively. The symptoms are dominated by muscle atrophy and muscle weakness, with upper limb dysfunction, gait disturbance, dysarthria, dysphagia, and respiratory impairment appearing with the progression of illness, and with no sensory dysfunction or dysuria. As the mechanism of motor neuron death, excitatory amino acid hypothesis, free radical hypothesis, and viral infection hypothesis have been proposed.

Rilutek® (riluzole) was first approved by the United States (US) Food and Drug Administration (FDA) in December 1995. Riluzole is indicated to extend life or the time to mechanical ventilation for subjects with ALS and represents the baseline standard of pharmacological care. Additional care is provided to reduce symptomatic medical concerns. Survival of subjects with ALS has improved over time, mainly as a result of the improvement in the symptomatic care of ALS.<sup>7,8</sup>

Edaravone (MT-1186, MCI-186), developed by Mitsubishi Tanabe Pharma Corporation, is a free radical scavenger that reduces oxidative stress and slows the progression of ALS as estimated by the Revised ALS Functional Rating Scale (ALSFRS-R). The clinical development program was designed to evaluate functional changes in ALS versus placebo up to 24 weeks. The concomitant use of riluzole was permitted in both edaravone and placebo groups. Efficacy of edaravone has been demonstrated in definite or probable subjects with ALS diagnosed with El Escorial criteria. 9,10,11,12 Higher relative quality of life has been demonstrated in subjects receiving edaravone compared to the placebo group, and these differences were maintained up to 48 weeks. 13 Evidence regarding the delay of some of the definite disease progression events (including death, disability of independent ambulation, loss of upper limb function, tracheotomy, use of respirator, use of tube feeding, and loss of useful speech) was also found at 48 weeks. 13 During the edaravone clinical development program, all fatal events, which occurred after respiratory failure, pneumonia or cardiac arrest, or serious adverse events (SAEs) such as gastrointestinal or respiratory disorders, were attributed or suspected to be attributed to disease progression. However, higher incidence of contusion, gait disturbance, headache, eczema, contact dermatitis, and glucosuria was reported in the edaravone group.<sup>14</sup> Most of the population of the clinical development

program of edaravone was Japanese. However, a pharmacokinetic (PK) analysis compared Japanese and Caucasian populations, and no differences were observed between them. 15

In 2015, edaravone was approved in Japan and South Korea (as Radicut®) as a therapeutic option to slow down the progression of the disease in subjects with ALS. This was followed by approval (as Radicava®) by the US FDA in 2017 and the Health Canada (as Radicava<sup>TM</sup>) in 2018. It was approved in Switzerland and China in 2019, Indonesia in 2020, and Thailand in 2021.

Edaravone oral suspension for the treatment of ALS was approved in the United States in May 2022 under the trade name RADICAVA ORS®.

# 6.1.1 Known Potential Benefits and Previous Experience with the Oral Formulation

# 6.1.1.1 Benefits of Edaravone

Edaravone was first approved in Japan in 2001 for acute ischemic stroke (AIS). The approved dosing regimen for AIS is 30 mg administered as an intravenous (IV) infusion over 30 minutes twice daily up to 14 days. Clinical and nonclinical data collected to date indicate that edaravone is well tolerated and has a favorable benefit to risk ratio.

Although studies of many drugs have been conducted, no effective therapy to cure ALS has currently been established. Riluzole modestly extends life or the time to mechanical ventilation for subjects with ALS. Current ALS treatment focuses on symptomatic treatment and therapy, such as gastrostomy for dysphagia and use of a respirator for dyspnea.

Radicut (edaravone) injection was approved by Japanese Pharmaceuticals and Medical Devices Agency on 26 June 2015 and Radicava (edaravone) injection was approved by the US FDA on 05 May2017 for the treatment of ALS as an IV formulation containing 30 mg MCI-186 in 100 mL solution. Radicava was also approved in South Korea (2015), Canada (2018), Switzerland, China (2019), Indonesia (2020), and Thailand (2021). The approved dosage is a 60 mg IV infusion administered over 60 minutes following 4-week dosing cycles:

- Initial treatment cycle: daily dosing for 14 days followed by a 14-day drug-free period
- Subsequent treatment cycles: daily dosing for 10 days out of 14-day periods, followed by 14-day drug-free periods

As the Sponsor recognized long-term frequent IV infusion might be inconvenient for certain subjects and caregivers, the Sponsor started development of an oral formulation of edaravone for ease of administration for subjects and caregivers. Since subjects with ALS may develop swallowing difficulties, an oral suspension formulation of appropriate consistency and viscosity is proposed for clinical studies and ultimately as a to-be-marketed product.

Two-week toxicology studies in rodents (rats) and non-rodents (dogs) using the edaravone oral suspension were conducted in compliance with Good Laboratory Practice. The results demonstrated no new safety findings up to 300 mg/kg/day compared to safety events observed from previously reported IV administered toxicology studies. More recently, a

39-week toxicology study in non-rodents (dogs), and a 26-week study in rodents (rats) were completed. Findings observed in studies with rats at the top dose (250 mg/kg) included extramedullary hematopoiesis in the spleen and acinar cell hypertrophy in the submandibular gland, while the top dose in dogs (300 mg/kg) included abnormal gait, loss of patella reflex, vacuolation in the dorsal funicle of the white matter in the spinal cord, and vacuolation and atrophy of nerve fibers in the sciatic nerve.

# 6.1.1.2 Previous Clinical Experience with Oral Edaravone

# Study MT-1186-J01

Study MT-1186-J01 was a Phase 1 study that evaluated the PK, safety, and tolerability of oral edaravone in healthy adult males following single and multiple doses. In each cohort of the single ascending dose sub-study (Part 1), 6 subjects received edaravone (30 mg to 300 mg) and 2 subjects received placebo. Subjects in Cohorts 1 to 6 were Japanese and subjects in Cohort 7 were Caucasian. In the multiple ascending dose sub-study (Part 2), each cohort had 6 subjects on edaravone (120 mg and 200 mg) and 3 subjects on placebo.

Following increasing oral doses, edaravone was well absorbed with time to maximum concentration ( $t_{max}$ ) values of 0.29-0.75 hr. The maximum concentration ( $C_{max}$ ) and area under the concentration-time curve (AUC) of edaravone increased to a more than proportional degree within the dose range of 30 mg to 300 mg. The  $C_{max}$  and AUC after the administration of 120 mg oral edaravone suspension exceeded those of the 60 mg/60 minute IV marketed infusion. Approximately 105 mg of oral edaravone appears to be sufficient to achieve similar  $C_{max}$  and AUC values compared to those after 60 mg/60 minute IV marketed infusion. There was no statistically significant difference in the PK profile of edaravone between healthy Japanese and Caucasian subjects.

A significant food effect was observed following the oral administration of MT-1186. In the fed condition, MT-1186  $C_{max}$  was reduced by approximately 80% and AUC was reduced by approximately 60% compared to those in the fasted condition. This result indicates that oral MT-1186 suspension should not be administered with a meal.

When edaravone (120 mg and 200 mg) was administered orally once daily (30 minutes before breakfast) for 5 days, no accumulations in C<sub>max</sub> and AUC were observed for edaravone.

### Study MT-1186-J02

# Part 1: Drug-Drug Interaction Study

Based on the results from in vitro drug-drug interaction (DDI) studies conducted according to the FDA Guideline, the Sponsor has decided that a cytochrome P450 (CYP) 3A4induction study, a breast cancer resistance protein (BCRP) inhibition study, and an organic anion transporter (OAT) 3 inhibition study are necessary in humans, and other in vivo DDI studies are deemed unnecessary.

PK profiles after single doses of 50 mg sildenafil (CYP3A4 substrate), 10 mg rosuvastatin (BCRP substrate), and 40 mg furosemide (OAT3 substrate) were compared to PK profiles

after single doses of those drugs in combination with 120 mg of oral edaravone suspension. The oral dosing of edaravone at a dose of 120 mg did not have an effect on the PK of each substrate.

# Part 2: Preliminary Regimen-Finding Study

In Study MT-1186-J01, significant reductions in  $C_{max}$  and AUC values were observed under fed conditions. Therefore, in Study MT-1186-J02, the timing of administration of edaravone relative to meals (1 hour before or 4 hours after a high-fat meal) was preliminarily investigated in Japanese healthy subjects. Dosing of edaravone 1 hour prior to a high-fat meal showed slightly lower  $C_{max}$ , with  $t_{max}$  before 1 hour resulting in a slightly lower AUC compared to  $C_{max}$  and AUC in the fasted condition. However, these are likely due to variability in PK data rather than a food effect because the food conditions until 1 hour after dosing were the same between the fasted cohort and the 1 hour prior to meal cohort. Dosing of edaravone 4 hours after a high-fat meal reduced  $C_{max}$  to 55.9% and AUC from time 0 to 24 hours (AUC<sub>0-24h</sub>) to 76.3%, compared to that previously observed under fasting conditions.

# Study MT-1186-J03

Based on PK data obtained from previous studies in healthy volunteers, an oral suspension dose of 105 mg of edaravone is estimated to show an equivalent mean AUC compared to that of the 60 mg/60 minute IV infusion regimen. Therefore, PK profiles of 105 mg of oral edaravone suspension were compared to those of the 60 mg/60 minute IV infusion regimen as the approved dose in a planned confirmatory PK study in a crossover study design in Japanese healthy subjects (planned number of subjects was n = 42).

This study demonstrated that the 105 mg oral suspension has an equivalent area under the concentration-time curve from time 0 extrapolated to infinity (AUC<sub>0- $\infty$ </sub>) to the approved 60 mg/60 minute IV infusion regimen dose (geometric mean ratio [90% confidence interval (CI)]: 0.977 [0.917, 1.041]). Geometric mean ratio of  $C_{max}$  of 105 mg oral suspension compared to 60 mg/60 min IV infusion regimen was also within the bioequivalence range, but the upper limit of 90% CI exceeded 1.25 (geometric mean ratio [90% CI]: 1.217 [1.090, 1.359]).

The AUC<sub>0- $\infty$ </sub> of sulfate and glucuronide after oral dosing of 105 mg MT-1186 were 1.3 and 1.7 times higher than that of IV 60 mg/60 minute infusion regimen, respectively.

### Study MT-1186-A01

This was a global, multicenter, open-label, Phase 3 study that evaluated the long-term safety and tolerability of oral edaravone in patients with ALS. The primary safety analysis was assessed at Weeks 24 and 48. Patients received a 105-mg dose of oral edaravone administered in treatment cycles that replicated the dosing of IV edaravone.

The safety analysis of the study included 185 patients. The most common treatment-emergent adverse events (TEAEs) reported by  $\geq$ 5% of patients were fall (22.2%), muscular weakness (21.1%), constipation (17.8%), dyspnea (10.8%), dysphagia (10.3%), and back pain (10.3%). There were no serious TEAEs, TEAEs leading to death, or TEAEs related to study drug. This

study demonstrated that oral edaravone was generally safe and well tolerated during 48 weeks of treatment with no new safety concerns identified.

# Study MT-1186-J04

This was a clinical pharmacology study conducted to evaluate the PK of oral edaravone in subjects with ALS who were living independently (n=9). The study compared the differences in the PK of ALS patients versus the PK in normal healthy volunteers. No significant differences in the PK profile of edaravone were observed between healthy subjects and ALS patients.

# Study MT-1186-J05

This clinical pharmacology study was conducted to evaluate the PK of oral edaravone in ALS subjects when administered via a percutaneous endoscopic gastrostomy (PEG) tube. This study evaluated the difference in PK between edaravone suspension administered through a PEG tube versus historic oral administration in ALS subjects (Study J04) without a PEG tube. Preliminary data obtained from 6 completing ALS patients where oral edaravone suspension was administered via a PEG tube yielded exposures (AUC and C<sub>max</sub>) that were slightly higher (~30%) than noted previously in Study J04. The range of exposures noted in Study J05 was within the range previously observed in normal Japanese subjects and ALS subjects without a PEG tube. This modest increase in exposure following administration of the suspension through a PEG tube is not considered clinically significant.

# **Study MT-1186-J06**

The appropriate timings of oral administration relative to the timing and different types of meals were further investigated in this study. The results demonstrated that the following food conditions had little effect on the PK of MT-1186: intake of a high-fat meal (1000 calories, 50% fat) 8 hours before dose, intake of a low-fat (normal) meal (400 calories, 25% fat) 4 hours before dose, or intake of a caloric supplement (e.g., ENSURE LIQUID) 2 hours before dose.

# MT-1186-Z-101

This randomized, open-label, crossover, single dose clinical pharmacology study was conducted in 36 healthy volunteers to assess the comparative bioavailability of oral edaravone when administered via nasogastric tube (a surrogate for PEG/radiologically inserted gastrostomy [RIG] administration) compared to oral administration. PK data obtained from 36 subjects showed that both C<sub>max</sub> and AUC fell within equivalence criteria. These data indicate that oral edaravone can be administered orally and via PEG/RIG without any need for dose adjustment.
## 7 STUDY OBJECTIVES, ENDPOINTS, AND HYPOTHESES

## 7.1 Study Objectives

## 7.1.1 Primary Objective

- To evaluate and compare the efficacy of the following 2 dosing regimens of oral edaravone in subjects with ALS, based on the time from the randomization date in Study MT-1186-A02 to at least a 12-point decrease in ALSFRS-R or death, whichever happens first, over the course of the study or until oral edaravone is commercially available in that country:
  - Oral edaravone 105 mg administered once daily
  - Oral edaravone 105 mg administered for 10 days followed by placebo for 18 days (regimen denoted as on/off).

## 7.1.2 Secondary Objective

• To evaluate the safety and tolerability of oral edaravone at a dose of 105 mg once daily compared to oral edaravone at a dose of 105 mg including placebo (regimen denoted as on/off) in subjects with ALS over the course of the study or until oral edaravone is commercially available in that country.

## 7.2 Study Endpoints

## 7.2.1 Primary Efficacy Endpoint

• Time from the randomization date in Study MT-1186-A02 to at least a 12-point decrease in ALSFRS-R or death, whichever happens first.

## 7.2.2 Secondary Efficacy Endpoints

- The Combined Assessment of Function and Survival (CAFS) score at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04
- Change in the ALS Assessment Questionnaire 40 score at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04
- Change in ALSFRS-R score at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04
- Time from the randomization date in Study MT-1186-A02 to death, tracheostomy, or permanent assisted mechanical ventilation (≥23 hours/day)
- Time from the randomization date in Study MT-1186-A02 to death or permanent assisted mechanical ventilation (≥23 hours/day)
- Time from the randomization date in Study MT-1186-A02 to death

## 7.2.3 Exploratory Efficacy Endpoints

- Change in percent slow vital capacity (SVC) at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04
- Change in body weight at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04
- King's ALS Clinical Stage derived from ALSFRS-R score and death at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04

## 7.2.4 Safety Endpoints

- Adverse events (AEs), adverse drug reactions, and TEAEs (e.g., grade, incidence, severity)
- Physical examination
- 12-lead electrocardiogram (ECG) parameters
- Vital signs (heart rate, respiratory rate, sitting systolic and diastolic blood pressure, and axillary, oral, temporal [skin-based], or tympanic body temperature)
- Laboratory safety assessments (e.g., hematology, chemistry, and urinalysis)
- Columbia-Suicide Severity Rating Scale (C-SSRS)

## 7.2.5 Hypothesis

Edaravone is expected to slow disease progression based on ALSFRS-R score and increase survival time.

## 8 STUDY DESIGN

## 8.1 Overall Study Design

This is a Phase 3b, multicenter, double-blind, parallel group, randomized extension study that will evaluate the efficacy and safety of 2 treatment regimens of edaravone for an additional period of up to 48 weeks following Study MT-1186-A02 in subjects with ALS as follows:

- Group 1: Oral edaravone 105 mg dose once daily in each 28-day cycle for up to 48 weeks or until the drug is commercially available in that country.
- Group 2: Oral edaravone 105 mg dose for 10 days followed by 18-day placebo (regimen denoted as on/off) in each 28-day cycle for up to 48 weeks or until the drug is commercially available in that country.

Subjects who meet study MT-1186-A04 eligibility criteria, will continue in the same treatment group/regimen that they were in during Study MT-1186-A02.

A schedule of assessment of all study procedures is provided in Table 1.

The Week 48 study procedures from Study MT-1186-A02 will be used as the screening/entry criteria for Study MT-1186-A04, followed by a treatment period of up to an additional 48 weeks or until oral edaravone is commercially available in each country, whichever time period is shorter, and a safety follow-up period of 2 weeks.

During the conduct of Study MT-1186-A04, the dose of edaravone may be adjusted or the study may be stopped based on the interim futility or final analyses performed for Study MT-1186-A02, taking into consideration the benefit and risk balance. However, unless any significant safety issue is found based on these 2 analyses, the same regimen will be kept while maintaining the blind conditions for all site-facing personnel and all personnel directly involved with the conduct of the study.

Concomitant use of riluzole is permitted throughout the course of the study when the dose and regimen remain unchanged from the screening visit evaluation of ALSFRS-R of Study MT-1186-A02 through the end-of-treatment (EOT) or early termination (ET) of Study MT-1186-A04. Dose reduction, dose interruption, or discontinuation due to the onset of AEs, progression of dysphagia, or gastrostomy while on oral edaravone 105 mg are allowed. The use of AMX0035 will be allowed for patients in the event that it becomes commercially available via prescription in their respective country. AMX0035 should be taken at least 1 hour after MT-1186/oral edaravone dosing.

EOT assessments will occur at Week 48 (Visit 5).

For subjects who complete the double-blind treatment period, a safety follow-up telephone visit will occur at Week 50 (Visit 6).

Subjects will be allowed to change from oral administration to PEG/RIG tube administration during the study.

Subjects who discontinue early from the study will complete the procedures listed at Week 48 (refer to Table 1 for further information) within 7 days of discontinuation. Site staff should also follow up via phone call at all remaining visits to complete the assessment for time to tracheostomy or permanent assisted mechanical ventilation, or death.

Further details can be found in the Study Schema (Figure 1).

## 8.2 Rationale for Study Design

The rationale for the study design is to assess the long-term efficacy of oral edaravone in subjects with ALS at doses of 105 mg administered once daily compared to a dose of edaravone at 105 mg administered for 10 days, followed by placebo for 18 days in each cycle (regimen denoted as on/off) for a total treatment duration of up to 48 weeks following Study MT-1186-A02 (2 years total exposure).

#### 8.2.1 Risk/Benefit Assessment

Edaravone has been evaluated in six Phase 1 studies in healthy subjects in Japan and Europe and has been evaluated in other clinical studies, including ALS, as follows:

- 8 clinical studies in AIS subjects in Japan and Europe with IV edaravone
- 3 clinical studies in subarachnoid hemorrhage subjects in Japan with IV edaravone
- 5 clinical studies in ALS in Japan with IV edaravone
- 7 clinical studies with oral edaravone

The treatment of AIS and ALS in Japan states that IV edaravone (MCI-186) is contraindicated in subjects with severe renal impairment and should be administered with care in subjects with hepatic impairment. Conversely, there are no contraindications or warnings to subjects with renal or hepatic impairment in the United States Prescribing Information (USPI) for treatment of ALS in the US.

In the USPI (IV edaravone) Warnings and Precautions section, hypersensitivity reactions (redness, wheals, and erythema multiforme) and cases of anaphylaxis (urticaria, decreased blood pressure, and dyspnea) have been reported in spontaneous post-marketing reports with edaravone. Edaravone contains sodium bisulfite, a sulfite that may cause allergic type reactions, including anaphylactic symptoms and life-threatening or less severe asthmatic episodes in susceptible people. The overall prevalence of sulfite sensitivity in the general population is unknown. Sulfite sensitivity occurs more frequently in asthmatic people.

In the USPI (IV edaravone) adverse reactions section, the most common adverse reactions observed during clinical studies were contusion, gait disturbance, headache, dermatitis, eczema, respiratory failure, respiratory disorder, hypoxia, glycosuria, and tinea infection.

Risk related to Coronavirus disease 2019 (COVID-19) was also assessed. Edaravone is not known to alter immune function. However, there may be additional risk to participants due to exposure to COVID-19 during study related visits (dependent on the country/region conditions). Subjects will be encouraged to observe social distancing, wear face masks/coverings, and avoid social gatherings during the conduct of the clinical trial and site

visits if COVID-19 is prevalent. Additionally, the Sponsor will monitor country conditions and prepare contingency plans for COVID-19 related restrictions that may prevent site visits.

#### 8.2.2 Rationale for Dose Selection

Study MT-1186-J03 results have demonstrated that a 105 mg oral suspension has an equivalent AUC to the approved 60 mg/60 min IV dose (geometric mean ratio [90% CI]: 0.977 [0.917, 1.041]). The geometric mean ratio of  $C_{max}$  of 105 mg oral suspension compared to 60 mg/60 min IV was also within bioequivalence range, but the upper limit of 90% CI exceeded 1.25 (geometric mean ratio [90% CI]: 1.217 [1.090, 1.359]). Therefore, the dose in this protocol has been set at 105 mg.

The currently marketed IV dosing regimen is the on/off regimen, with patients taking medication for 10 out of 14 days followed by a 14-day medication-free period, resulting in 28-day cycles. This dosing regimen was based on the treatment regimen of edaravone indicated for AIS. The daily dose and the overall design of this study was chosen in conjunction with the FDA as a post-marketing commitment, in hopes of providing patients with a more convenient dosing regimen and the potential benefit of daily (continuous) dosing.

## 8.2.3 Independent Data Monitoring Committee

An Independent Data Monitoring Committee (IDMC) composed of experts in the management of subjects with the disease under study and a biostatistician will review unblinded interim safety data with risk-benefit periodically, at predefined intervals, during the study. Any such reviews of study data will be undertaken in accordance with predefined rules and procedures. These rules will be implemented to ensure that access to details of the study blind, and to unblinded data, is carefully controlled. A charter will guide the timing of reviews; communications between the IDMC, the Investigators, and the Sponsor; and stopping rules for the study. In general, the IDMC will advise the Sponsor regarding possible changes to the protocol or study procedures to protect the subjects enrolled in the study.

The specific details about the IDMC will be included in an IDMC charter.

## 9 SELECTION AND WITHDRAWAL OF SUBJECTS

## 9.1 Number of Subjects

Approximately 300 subjects (150 subjects per dosing group) who have successfully completed Study MT-1186-A02 (completion through Week 48 [Visit 15]) and who meet Study MT-1186-A04 eligibility criteria will be enrolled.

#### 9.2 Recruitment Methods

Subjects will be recruited upon completion of the MT-1186-A02 study. Only subjects who are eligible for the study based upon their Week 48 procedures from the MT-1186-A02 study will be enrolled.

#### 9.3 Inclusion Criteria

Subjects who meet all of the following criteria will be considered eligible to participate in Study MT-1186-A04:

- 1. Subjects or their legally authorized representative (LAR) must provide a signed and dated ICF to participate in the study.
- 2. Subjects must be able (in the judgment of the Investigator) to understand the nature of the study and all risks involved with participation in the study.
- 3. Subjects must be willing to cooperate and comply with all protocol restrictions and requirements.
- 4. Subjects must have successfully completed all Study MT-1186-A02 visits and have been compliant with study drug.

## 9.4 Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from the study:

- 1. Subjects of childbearing potential unwilling to use an acceptable method of contraception from the Day 1/screening visit until 3 months after the last dose of study medication. Subjects who are sexually active who do not agree to use contraception during the study period. Refer to Appendix 3 for additional contraceptive information.
- 2. Subjects who are female, of childbearing potential, and pregnant (a positive pregnancy test) or lactating at the Day 1/screening visit.
- 3. Subjects who have a significant risk of suicide. Subjects with any suicidal behavior or suicidal ideation of type 4 (active suicidal ideation with some intent to act, without a specific plan) or type 5 (active suicidal ideation with specific plan and intent) based on the C-SSRS at Week 48 of Study MT-1186-A02.
- 4. Subjects who are not eligible to continue in the study, as judged by the Investigator in conjunction with the MTDA medical monitor.
- 5. Subjects who are unable to take their medications orally or through a PEG/RIG tube.

#### 9.5 Screen Failures

If a subject has not met all eligibility criteria at the beginning of the treatment period, the subject will be registered as a screen fail and cannot be enrolled into the study.

## 9.6 Withdrawal of Individual Subjects

A subject will be withdrawn from the study if the subject meets any of the following criteria:

- The subject is lost to follow-up
- The subject requests to be withdrawn from the study
- The subject has been found to be ineligible for participation in the study
- The Investigator (or sub-investigator) judges continuation of the study to be difficult due to AEs (e.g., hypersensitivity reactions)
- The subject is pregnant
- The subject requires tracheostomy
- The subject requires permanent assisted mechanical ventilation (≥23 hours/day)
- The Investigator (or sub-investigator) judges continuation of the study to be inappropriate due to exacerbation of the primary disease
- The subject has significant hepatic abnormalities:
  - Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >8 × upper limit of normal (ULN) OR
  - Persistent ALT or AST >5 × ULN OR
  - ALT or AST  $>3 \times$  ULN with concomitant bilirubin  $>2 \times$  ULN
  - Symptoms consistent with liver dysfunction (e.g., fatigue, nausea, vomiting, abdominal pain/tenderness, fever, rash, eosinophilia >5%) with concomitant ALT or AST >3 × ULN
  - Note: subjects meeting these criteria do not require withdrawal if alternative etiology is unequivocally identified on discussion with the Sponsor Medical Monitor
- Noncompliance (i.e., the subject misses more than 20% of doses in 2 consecutive dosing cycles [after consultation with MTDA or designee]).

If a subject is withdrawn prematurely from the study, the date the subject is withdrawn from the study and the reason for withdrawal will be recorded in the electronic case report form (eCRF).

If a subject drops out of the study at any time, the reason for discontinuation must be fully documented in the source documents and the eCRF. The investigator site personnel will document the AEs and any other assessments in the source documents and will make every effort to complete all required ET assessments. Study sites must follow-up with phone calls to assess for events at Weeks 12, 24, 36, and 48.

Subjects who withdraw due to liver dysfunction should be followed until resolution and assessed for alternative etiologies.

Subjects who are withdrawn from the study following enrollment may not re-enter the study.

The study may be terminated by the Sponsor at any time upon becoming aware of data that could compromise the safety and/or well-being of the subjects or for any other reason it deems appropriate.

## 10 STUDY PLAN

## 10.1 Description of Study Periods

Refer to Table 1 for an outline of procedures required at each study period and/or visit.

Prior to performing any study procedures, the Investigator (or designated personnel) will ensure that the subject is given full and adequate oral and written information about the study and the subject must sign the ICF, as described in Section 18.2.1.

#### 10.1.1 Double-blind Treatment Period

Subjects who successfully completed the Week 48 study procedures from Study MT-1186-A02 will remain at the study clinic, and inclusion and exclusion criteria will be reviewed against those Week 48 results to confirm eligibility. Eligible subjects will then be enrolled in Study MT-1186-A04, and dosing will begin on Day 1 (Visit 1) and will continue in the study for up to 48 weeks.

Study visits will occur onsite, in the patient home, or via a telephone call per the Schedule of Assessments (Table 1).

## 10.1.2 Optional Open Label Treatment Period

If, based on the results of Study MT-1186-A02 or recommendations of the IDMC, either the daily dose regimen or the on/off regimen are demonstrated to be safer or more effective, the study will convert to an open-label treatment study and all remaining patients will be converted to the optimal arm at the earliest possible visit.

## 10.1.3 End-of-Treatment/Early Termination Period

The EOT visit will occur at Week 48.

For subjects who terminate early from the study, assessments should be performed per the Schedule of Assessments (Table 1) as close to the termination date as possible. The ALSFRS-R should be administered by the same Investigator or sub-investigator throughout the study whenever possible, including any ETs.

Any unresolved AE or SAE will be followed up according to Section 15.8.

If a subject selects not to return to the clinical site for the ET Visit, the Investigator must make every effort to contact the subject to review all AEs. If a subject drops out of the study at any time, the reason for discontinuation must be fully documented in the source documents and the eCRF. The Investigator site personnel will document the AEs and any other assessments in the source documents and will make every effort to complete all required ET assessments. For all subjects, Visit 5 (ET, Week 48) assessments should be performed, per the Schedule of Assessments (Table 1).

## 10.1.4 Safety Follow-up Period

A safety follow-up call (e.g., Week 50 [±7 days]) will be conducted for all subjects who complete the treatment period of the study.

## 10.1.5 End-of-Study Options

The EOT visit will occur at either Week 48, when the drug is commercially available in that country, if results from Study MT-1186-A02 dictate, or in the event the Sponsor discontinues the study.

#### 10.1.6 Unscheduled Visits

An unscheduled visit is defined as any visit to the Investigator site outside of the protocol-specified time points due to safety reasons or when a repeated measurement is required (e.g., obvious measurement errors, measuring device failure, confirmation of out-of-range results), or if a medication regimen change is required, where the subject is seen by study personnel.

Due to COVID-19 restrictions related to site visits, safety assessments such as routine blood sampling or other assessments may be performed in the subject's home at the discretion of the Investigator and based upon the site's abilities, including the performance of complete study visits or questionnaires via telephone. All assessments performed during the visits will be recorded in the eCRF.

## 11 STUDY PROCEDURES

All subjects must sign and date the IRB/IEC-approved ICF before any study-specific procedures are performed. Refer to Section 18.2.1 for further details.

## 11.1 Concomitant Medications

Concomitant medication is defined as any medication, other than the study drug, that is taken from the screening visit in Study MT-1186-A02 to the MT-1186-A04 end-of-study (EOS) visit, including prescription, herbal, and over-the-counter medications. All concomitant medications taken while the subject is participating in the study will be recorded in the eCRF (including riluzole and AMX0035).

#### 11.2 Prohibited Concomitant Medications

Concomitant use of the following drugs and any other investigational products will be prohibited from the Day 1/screening visit through the end of Week 50 or the time of discontinuation:

- Masitinib
- Ropinirole
- Tauroursodeoxycholic acid (except in the form of AMX0035)
- Phenylbutyrate (except in the form of AMX0035)

## 11.3 Permitted Concomitant Medications

Concomitant use of riluzole will be permitted when the dose and regimen remain unchanged from the screening visit evaluation of ALSFRS-R of Study MT-1186-A02 through the EOT/ET of Study MT-1186-A04. Dose reduction, dose interruption, or discontinuation due to the onset of AEs, progression of dysphagia, or gastrostomy while on oral edaravone 105 mg are allowed. New or additional use of AMX0035 will be allowed for patients once it becomes commercially available in their respective country. AMX0035 should be taken at least 1 hour after MT-1186/oral edaravone dosing. Use of riluzole and AMX0035 will be recorded in the CRF.

For subjects who take a supplemental vitamin B6, it is recommended to take the smallest feasible therapeutic dose at bedtime.

COVID-19 and other vaccines that have received emergency use authorization or approval are allowed. At a minimum, the following must be documented in the concomitant medication section of the eCRF: the type of vaccine, the manufacturer of the vaccine, and the date(s) the subject received the vaccine.

## 12 EFFICACY ASSESSMENTS

## 12.1 Primary Efficacy Assessment

## 12.1.1 ALS Functional Rating Scale

The Investigator (or sub-investigator) will attend a certified rater training for ALSFRS-R to ensure consistent and accurate ratings.

The Investigator (or sub-investigator) will evaluate subjects using the ALSFRS-R and rater scores will be collected at the time points described in Table 1.

Appendix 2 is an example of a questionnaire used to measure the impact of ALS that is evaluated by the Investigator. The scale measures the subject's physical function across 12 activities of daily living. The date of the evaluation along with the results will be recorded in the eCRF. With respect to "4 Handwriting" and "5 Eating motion," the results for the dominant hand (the hand used in daily life at the time of Day 1 of Study MT-1186-A02) will be recorded in the eCRF.

## 12.2 Secondary Efficacy Assessment

## 12.2.1 Combined Assessment of Function and Survival Score

The CAFS score will be calculated by the Sponsor to compare individual subjects to all other subjects using ALSFRS-R and date of death event as described in Table 1.

## 12.2.2 Time to Death, Tracheostomy, or Permanent Assisted Ventilation

The Investigator (or sub-investigator) will investigate the presence or absence of the following events from the randomization date in Study MT-1186-A02 through EOT/ET in Study MT-1186-A04:

- Time (days) to death
- Time (days) to tracheostomy
- Time (days) to permanent assisted mechanical ventilation (≥23 hours/day)

If any of the events are present, the following will be investigated and recorded in the eCRF: the date of the event and EOS date. When a subject discontinues from the study, study sites must follow-up with phone calls at the time points described in Table 1. The evaluation results, together with the dates of the evaluation, will be recorded in the eCRF.

## 12.3 Exploratory Efficacy Assessment

### 12.3.1 Slow Vital Capacity

Evaluators need to be trained and appropriately qualified to perform this test. Certified calibration free spirometry equipment will be provided by a central spirometry provider, which will meet core American Thoracic Society (ATS)/European Respiratory Society (ERS)

criteria for reproducibility. SVC measurements will be conducted in the clinic at around the same time of day, when possible, with the subject sitting in an upright position. Subjects should make at least 3 attempts to generate acceptable and reproducible SVC data per ATS/ERS guidelines. If subjects cannot complete all 3 attempts due to disease progression or other reasons, it will not be considered a protocol deviation. The best value will be selected and will be recorded in the eCRF. A quality review of the data generated will also be conducted by a central over-read specialist, and feedback will be provided to the site.

## 12.3.2 Body Weight

Body weight will be measured and recorded in pounds or kilograms.

## 12.3.3 King's ALS Clinical Stage Derived from ALSFRS-R Score and Death Event

The King's ALS clinical stage will be calculated by the Sponsor at each visit using ALSFRS-R and event of death.

## 13 SAFETY ASSESSMENTS

## 13.1 Physical Examination

A full physical examination will consist of an assessment of major body parts and systems: abdominal, cardiovascular, general appearance, head, eyes, ears/nose/throat, lymph nodes, musculoskeletal, neck, neurological, dermatological, respiratory, and other.

A routine physical examination will consist of an assessment of the following body parts and systems: abdominal, cardiovascular, general appearance, respiratory, neurological, and other.

Abnormalities of clinical significance will be reported as AEs.

## 13.2 Vital Signs

The following measurements will be performed: sitting systolic and diastolic blood pressure, heart rate (e.g., beats per minute), respiratory rate, and axillary, oral, temporal (skin-based), or tympanic body temperature (e.g., Celsius); the same method is to be used throughout the study. Subjects must be in a sitting position in a rested and calm state for at least 5 minutes before blood pressure assessments are conducted. The position selected for a subject should be the same that is used throughout the study and documented in the eCRF.

The Investigator will perform an overall evaluation for safety purposes, and the recording will be reported as 'normal', 'abnormal clinically significant (CS)', or 'abnormal not clinically significant (NCS)'.

Abnormalities of clinical significance will be reported as AEs. Repeat measurements will be performed if needed.

## 13.3 Body Weight

Body weight will be measured and recorded in pounds or kilograms, at time points mentioned in Table 1.

## 13.4 12-lead Electrocardiogram

A 12-lead ECG will be performed after the subject has rested for at least 5 minutes in a supine position. The ECG must include the following measurements: R wave to R wave (RR) interval, heart rate, QRS, and QT. If available, corrected QT interval by Bazett (QTcB), and corrected QT interval by Fridericia (QTcF) should also be recorded. The Investigator will perform an overall evaluation of the ECG for safety purposes and the recording will be reported as 'normal', 'abnormal CS', or 'abnormal NCS'. Abnormalities of clinical significance will be reported as AEs. Repeat measurements will be performed if needed.

## 13.5 Clinical Laboratory Tests

Blood will be drawn at assigned time points for laboratory assessment (refer to Table 1 for further details).

As a guideline, the volume of blood to be sampled per time point will be approximately 10 mL, and the volume of the urine aliquot to be sampled per time point will be approximately 15 to 20 mL.

## 13.5.1 Hematology

Red blood cell count, hemoglobin, hematocrit value, white blood cell (WBC) count including differential, and platelet count.

## 13.5.2 Blood Chemistry

Albumin, total protein, AST, ALT, lactate dehydrogenase, alkaline phosphatase, c-reactive protein, total bilirubin, direct bilirubin, creatine kinase, total cholesterol, triglycerides, blood urea nitrogen, bicarbonate, serum glucose, serum creatinine level, uric acid, sodium, potassium, chloride, calcium, cystatin C, and vitamin B6 will be measured at the time points described in Table 1.

## 13.5.3 Urinalysis (Qualitative)

Protein, glucose, occult blood, WBCs, urobilinogen, and bilirubin will be measured at the time points described in Table 1.

## 13.5.4 Pregnancy Test

For female subjects of childbearing potential only, urine beta-human chorionic gonadotropin test and serum beta-human chorionic gonadotropin level will be conducted as per Table 1. If a subject is confirmed to be pregnant, the subject will be excluded/terminated from the clinical study.

## 13.6 Columbia-Suicide Severity Rating Scale (C-SSRS)

Appropriately trained site personnel will attend a certified rater training for the C-SSRS, to ensure consistent and accurate ratings.

The C-SSRS is an instrument that captures the occurrence, severity, and frequency of suicide-related ideations and behaviors during the assessment period. At each visit, the C-SSRS will be compared against the last visit. The C-SSRS must be administered by appropriately trained site personnel. Suicidal ideation is classified on a 5-item scale: 1 (wish to be dead), 2 (nonspecific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active suicidal ideation with some intent to act, without specific plan), and 5 (active suicidal ideation with specific plan and intent). The C-SSRS also captures information about the intensity of ideation, specifically the frequency, duration, controllability, deterrents, and reasons for the most severe types of ideation. Suicidal behavior is classified on a 5-item scale: 0 (no suicidal behavior), 1 (preparatory acts or behavior), 2 (aborted attempt), 3 (interrupted attempt), and 4 (actual attempt). More than 1 classification can be selected provided they represent separate episodes. For actual attempts only, the actual or potential lethality is classified for the initial, most lethal, and most recent attempts. C-SSRS assessment examples are provided in Appendix 5.

## 14 STUDY DRUG TREATMENT

## 14.1 Investigational Medicinal Product

## 14.1.1 Drug Product

The Sponsor will provide edaravone oral suspension (21 mg/mL) and matching placebo in amber bottles, with adapters and oral syringes for each subject for the duration of their participation in the study. The suspension bottles will contain 1050 mg of edaravone or matching placebo for 10 days of dosing. The Investigator, a study nurse, or the hospital pharmacy will dispense a sufficient quantity of edaravone bottles and ancillary kits consistent with each subject's daily dosage requirement and study visits according to the protocol.

Before administration, subjects or caregivers must shake the bottle for at least 30 seconds and confirm no precipitation layer is on the bottom of bottle. Then, 5 mL of suspension must be taken using the syringe to administer 105 mg of edaravone or placebo.

## 14.1.2 Study Drug Supply

Edaravone and placebo multi-use bottles will be packaged, labeled, and released according to Good Manufacturing Practices. All labeling will comply with applicable regulatory requirements. The Sponsor will provide all required release documentation for the finished product before it is dispatched.

The Sponsor will provide the necessary documentation, such as a Certificate of Analysis or Quality Control release document.

## 14.1.3 Formulation, Packaging, and Labeling

Documentation for edaravone or placebo bottles will include, but may not be limited to, the following information:

- Receipt date
- Description of drug package and drug product
- Lot/Batch/Code/other
- Expiration and manufacturing dates
- Investigational New Drug number
- Certificate of Compliance

## 14.1.4 Shipping, Receipt, Handling, and Storage

The Investigator or designee must maintain an accurate record of the shipment and dispensing of study drug in a Drug Accountability Log. Drug accountability will be noted by the field monitor during site visits and at the completion of the study. Subjects will be asked to return all unused study drug and packaging at each on-site clinic visit, at the end of the study, or at the time of study treatment discontinuation.

The investigational product should be stored at 2°C to 8°C (36°F to 46°F) in its original carton to protect it from light. Investigational product should not be frozen. Sites will be required to monitor temperature of the investigational product while on-site.

Subjects will be instructed to store the medication under refrigerated conditions and protected from light, according to the investigational medicinal product (IMP) clinical label.

## 14.1.5 Dispensing

Per interactive web response system (IWRS) instructions (at the baseline visit and each clinic visit), the Investigator or designee will provide the subject with the appropriate number of bottles of edaravone suspension for the administration treatment period. A record of the study medication dispensed to each subject will be maintained by the Investigator or designee in a Drug Accountability Log.

## 14.1.6 Study Medication Accountability

The pharmacist or designee must maintain an accurate record of the study medication shipment. During the study, the pharmacist will record the quantities of edaravone or placebo bottles dispensed on a Drug Accountability Log. The accountability (drug reconciliation) will be noted by the monitor during site visits and at the completion of the study. Edaravone, matching placebo, or ancillary kits are to be used only for this Protocol and not for any other purposes.

## 14.1.7 Disposal and Destruction

At study closeout, and as appropriate during the study, the Investigator/designee will return all used and unused study drug, packaging, kits, and a copy of the completed Drug Accountability Log to the Sponsor's designated vendor or to the address provided in the Investigator Binder at each site.

The study medication supply may be destroyed at the designated Sponsor facility or third party, as appropriate. Sites with documented drug destruction procedures and facilities may destroy drug on site after obtaining Sponsor approval and after completing drug accountability with the Sponsor's designated monitor.

## 14.2 Dosing of Edaravone or Placebo

All subjects enrolled will receive 1 of the following dose regimens:

Group 1: Oral edaravone 105 mg administered once daily for up to 48 weeks or until the drug is commercially available in that country. Each cycle is 28 days and begins with the first dose from the bottle ending in "01" and ends with the 28<sup>th</sup> dose from the last bottle in the kit.

Group 2: Oral edaravone 105 mg administered daily for 10 days followed by 18 days of placebo (regimen denoted as on/off) for up to 48 weeks or until the drug is commercially available in that country. Each cycle is 28 days and begins with the first dose from the bottle ending in "01" and ends with the 28<sup>th</sup> dose from the last bottle in the kit.

The dose of IMP should be taken after an overnight fast, and subjects must continue to fast at least 1 to 2 hours post-dose before the next meal (e.g., breakfast).

A description of edaravone or placebo study medication dispensed is provided in Table 3.

Table 3: Investigational Product

| Product Name: | Edaravone | Placebo |
|---|---|---|
| Dosage Form: | Oral suspension | Oral suspension |
| Unit Dose | 105 mg per 5 mL | Placebo |
| Route of Administration | Oral/PEG/RIG tube | Oral/PEG/RIG tube |
| Physical Description | Aqueous viscous suspension | Aqueous viscous suspension |
| Manufacturer | PCI Pharma Services (UK) | PCI Pharma Services (UK) |

## 14.3 Treatment Compliance

The prescribed dosage, timing, and mode of administration of study medication may not be changed except for PEG/RIG dosing as the subject's disease progresses. Subjects or caregivers will notify the study team of any medication doses missed. Subjects will be asked questions regarding study drug compliance and any departures from the intended regimen, including whether the subject has switched from oral dosing to PEG/RIG tube; the switch date must be recorded in the eCRF.

Study drug accountability and treatment compliance will be documented throughout the study period using study medication dispensing and return record logs.

Subjects will be asked to return all unused medication including empty and partially used medication. Study medication dispensed at the previous visit will be collected by the site and compliance will be assessed by counting the returned study medication bottles.

Non-compliance is defined as taking <80% or >120% of study medication during evaluation periods (cycle to cycle).

## 14.4 Subject Identification

Each subject will continue to be identified by the unique Subject Identifier that was assigned to them at the screening visit of Study MT-1186-A02.

The Subject Identifier will be used to reference the subject during the entire duration of the study. The Subject Identifier will be documented in the subject's source documents. The Subject Identifier will be recorded on study medication labels and other documentation.

A list identifying the subjects by their unique Subject Identifier will be kept in the Investigator Site File.

## 14.5 Procedures for Assigning Subjects to Treatment Groups

Enrollment will take place after confirmation of inclusion/exclusion criteria. Assignment of study medication will be performed through the interactive voice response system (IVRS)/IWRS, and subjects will continue in the same treatment group/regimen they were in during Study MT-1186-A02.

## 14.6 Maintenance of the Study Blind and Unblinding

During the double-blind treatment period, neither the subject nor the Investigator site personnel will know which treatment is being taken. Each subject will maintain their unique randomization number assigned from Study MT-1186-A02. The codes will only be accessible to authorized IVRS/IWRS users. Randomization numbers will be recorded in the eCRF.

The IVRS/IWRS should not be accessed to break the treatment code for reasons other than safety or in an emergency. Should the Investigator need to break the code for such reasons, he/she may access the IVRS/IWRS to obtain the treatment code and provide the system with the reason for breaking the blind. The Sponsor should be notified as soon as possible thereafter. The Investigator should promptly document and explain to the Sponsor any premature unblinding. If the blind is broken for any individual subject, the subject must be withdrawn from the study, and any procedures accompanying withdrawal should be performed.

The Sponsor and study team, except for the unblinded personnel involved with study safety assessments, will remain blinded to all subject randomization assignments throughout the duration of the double-blind treatment of the study until the interim data lock. Contract research organization (CRO) personnel will remain blinded during the double-blind treatment period.

An electronic list of randomization codes will be retrieved from IVRS/IWRS and transferred to the Sponsor after the interim database is locked for this study. No study personnel involved in the day-to-day conduct of the study will have access to unblinded data.

Edaravone and placebo are identical in appearance and will be packaged identically and suitably labeled to maintain the blind.

The handling of data that could potentially unblind the study will be defined in relevant study procedures documents (e.g., Blinding and Unblinding Plan or equivalent).

#### 14.7 Dose Adjustment Criteria

Dose adjustments of IMP will not be allowed. A dose adjustment may be initiated in the event that Study MT-1186-A02 results require all patients to convert to the other regimen/treatment.

## 15 ADVERSE EVENT MANAGEMENT

All AEs and SAEs will be recorded in the source documents. All AEs and SAEs that occur from the time written ICF is obtained until the end of the Safety Follow-up Period will be recorded in the eCRF. Even if an AE is assessed by the Investigator as not related to IMP, its occurrence must be recorded in the source documents and eCRF. AEs will be classified as 'treatment-emergent' if they arise following the administration of IMP or if a pre-dose AE increases in severity following dosing.

At each study visit, after the subject has had an opportunity to spontaneously mention any problems, the Investigator should inquire about the occurrence of AEs. The questioning should be open-ended and non-leading.

#### 15.1 Adverse Event

An AE is any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of an IMP, whether or not considered related to the IMP. Instances of aggravation of events (in terms of seriousness) are treated as new AEs.

#### 15.2 Serious Adverse Event

An SAE is defined as any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening
- Requires hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability or incapacity
- Is a congenital anomaly or birth defect
- Is an important medical event

Medical and scientific judgement should be exercised in deciding whether an AE is serious and whether expedited reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require medical or surgical intervention to prevent 1 of the other outcomes listed in the above definition. These should also be considered serious.

Examples of such events are invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse. These should also usually be considered serious.

The term 'life-threatening' refers to an event/reaction in which the subject was at risk of death at the time of the event/reaction; it does not refer to an event/reaction that hypothetically might have caused death if it were more severe.

Admission to a hospital as a new inpatient is deemed as meeting this criterion, even when the length of hospital stay was less than 24 hours. Transfer to other departments of the same hospital due to a newly emerged event during the hospitalization (e.g., transfer from the psychiatry ward to the internal medicine ward, from the internal medicine ward to the coronary intensive care unit, or from the neurology ward to the tuberculosis ward) is also counted as hospitalization.

SAEs will be recorded and reported as described in Section 15.7.

## 15.3 Severity of Adverse Events

The severity of AEs will be classified according to the following criteria:

Mild:

The event is transient and easily tolerated by the subject.

Moderate:

The event causes discomfort and interferes with the subject's general

condition.

Severe:

The event causes considerable interference with the subject's general condition

and may be incapacitating.

To ensure no confusion or misunderstanding of the difference between the terms 'serious' and 'severe', which are not synonymous, the following note of clarification is provided.

The term 'severe' is often used to describe the severity of a specific event (as in mild, moderate, or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as severe headache). This is not the same as 'serious', which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

## 15.4 Relationship of Adverse Events to Investigational Medicinal Product

The causal relationship of the AE to IMP will be determined as either 'reasonable possibility' or 'no reasonable possibility' defined as:

Reasonable Possibility – The relationship of the clinical event to the IMP makes a causal relationship possible, and other drugs, therapeutic interventions, or underlying conditions do not provide a sufficient explanation for the observed event.

No Reasonable Possibility – The relationship of the clinical event to the IMP makes a causal relationship unlikely, or other drugs, therapeutic interventions, or underlying conditions provide a sufficient explanation for the observed event.

## 15.5 Clinical Laboratory Abnormalities and Other Abnormal Assessments

The Investigator will exercise medical judgment in deciding whether abnormal laboratory test results are clinically significant. Laboratory abnormalities, which are CS, will be recorded as AEs or SAEs.

If an abnormal laboratory value or assessment is clearly related to a medically defined diagnosis or syndrome, the diagnosis or syndrome will be recorded on the AE form, not the individual laboratory values.

All 'abnormal, CS' laboratory results or assessments will be followed until they resolve (return to normal or baseline values) or stabilize, or until they are judged by the Investigator to be no longer CS. Repeat laboratory tests or measurements will be performed if needed.

## 15.6 Recording and Reporting of Adverse Events

All AEs, regardless of the relationship to IMP, occurring from the time written ICF is obtained from a subject until the end of the safety Follow-up Period or the withdrawal of the subject from the study will be recorded.

NOTE: Elective hospitalization or a procedure/surgery planned before subject enrollment in Study MT-1186-A02 for a pre-existing medical condition does not constitute an AE unless the underlying disease or condition worsens after signing the ICF.

All AEs will be recorded on an AE form in the eCRF. Reports should contain a description of the event, date and time of onset, date and time of resolution, severity, treatment required, relationship to IMP, action taken with the IMP, outcome, and whether the event is classified as serious.

The Investigator will evaluate the severity of the AEs (as defined in Section 15.3) and will assess the causality between the AEs and the IMP (as defined in Section 15.4).

Pre-existing illnesses/conditions, which started prior to the first dose of IMP, will not be considered AEs unless they worsen during the treatment period. Pre-existing illness/conditions will be recorded as medical history.

If the Investigator becomes aware of any new safety information, or any safety information that appears to be either study- or IMP-related after the final Follow-up Period, they must notify the Sponsor immediately.

## 15.7 Recording and Reporting of Serious Adverse Events

All SAEs occurring from the time written ICF is obtained from a subject until the end of the Safety Follow-up period or the withdrawal of the subject from the study must be reported to the Sponsor/CRO using the SAE Form in Clinical Study within 24 hours of the Investigator becoming aware of the SAE. All SAEs must also be entered in the AE section of the eCRF as soon as possible.

SAE reports should be completed as thoroughly as possible, including an assessment of causality. All such reports will identify subjects by unique code numbers assigned to the study participants, rather than by the subjects' names, personal identification numbers, or addresses.

The reporting contact for SAEs is as follows:

In case of any email problems, the SAE form can be sent to

via fax to:

Fax:

The Sponsor will comply with the applicable regulatory requirements related to the reporting of suspected unexpected serious adverse reactions (SUSARs) to the regulatory authorities and central IRBs. The Investigator will be responsible for informing the local IRBs of relevant safety information, including SUSARs, as per local laws and requirements.

## 15.8 Follow-up of Adverse Events

The Investigator should follow-up subjects with AEs/SAEs, until the event has resolved or stabilized, and any abnormal laboratory values have returned to normal or baseline values, or until there is a satisfactory explanation for the changes observed. In the case of death, if possible, a pathologist's full report should be supplied.

## 15.9 Pregnancy

If a female subject who has been exposed to the study medication becomes pregnant, the course and outcome of the pregnancy should be monitored and documented. Where possible, if a female partner of a male subject who has been exposed to the study medication becomes pregnant and the subject provides this information, then the pregnancy will be documented based on information provided by the subject.

A pregnancy that occurs in a subject who has been exposed to the study medication must be reported using the same timelines and contact details as an SAE (Section 15.2) by a paper *Pregnancy in a Clinical Study Notification Form*, although pregnancy alone will not be classified as an AE or SAE. If the outcome of the pregnancy or an event occurring during pregnancy involves an SAE (e.g., a congenital anomaly), then the *SAE in a Clinical Study Form* will also be completed.

Subjects who become pregnant while in the study should be withdrawn from treatment, as described in Section 9.6.

## 15.10 Reference Safety Information

The reference safety information for this clinical study is the edaravone Investigator's Brochure. 16

#### 15.11 Overdose

There is no known antidote for edaravone. Any signs or symptoms of a possible overdose will be treated supportively. In the case of an emergency, standard emergency procedures and supportive medical care will be given.

If the subject takes a dose that is greater or more frequent than that specified in the Protocol (with or without associated symptoms), this overdose is an AE and must be reported to the Sponsor or the designee on the AE eCRF.

If the overdose results in AEs that meet serious criteria, the SAE must be reported to the Sponsor or designee immediately or within 24 hours of awareness using the SAE Form in Clinical Study according to SAE reporting procedures (see Section 15.2).

## 16 DATA COLLECTION AND PROCESSING

#### 16.1 Data Collection

Subject data will be collected on individual eCRFs and will be substantiated by source documents (such as laboratory reports, medical records, or ECGs) at the Investigator site. All relevant data will be transcribed into the eCRF from source documents, entered into the study database directly from source documents, or transferred electronically to the study database. Where no printed or electronic source documents exist, data will be entered directly into the eCRF, electronic patient reported outcomes, and the bioanalytical databases (central laboratory) and the eCRF will be considered the source document.

Prior to the start of the study, the Investigator will complete a Delegation of Responsibility List. The Sponsor will provide training for completion of the eCRF. The eCRF will be completed according to guidelines provided by the Sponsor or its designee in writing, electronically, and/or verbally.

Completed eCRFs will be reviewed by the Study Monitor for the study to ensure data accuracy, completeness, and consistency. Any discrepancies found during the eCRF review or during data validation and/or quality assurance reviews of the data-by-data management or other functions are to be clarified by the Investigator (or his/her designated personnel).

The Investigator or designee must record all required subject data using the previously specified data collection method defined by the Sponsor. An explanation must be documented for any missing data. The Investigator must electronically sign and date a declaration in the eCRF attesting to his/her responsibility for the quality of all data recorded, and that the data represents a complete and accurate record of each subject's participation in the study. The data collected in the eCRF will be returned to the Sponsor, and an electronic copy will be retained by the Investigator.

## 16.2 Case Report Form

The Case Report Form will be presented in an electronic casebook comprising a series of electronic forms. The Subject Identifier should always be indicated and the date (and time, if applicable) of each assessment should be entered in the eCRF.

The eCRFs must be completed in a timely manner so that this does not delay the ongoing data validation, review, and quality control. The final, completed eCRF for each subject must be electronically signed and dated by the Investigator on the appropriate eCRF form to signify that he/she has reviewed the electronic casebook and certifies it to be complete and accurate.

The eCRF will feature a special means for correcting errors in the previously entered data. A complete audit trail of the original entries, changes and deletions, session dates and times, and the credentials of the eCRF user who performed the operation will be maintained by the system.

## 16.3 Data Processing

The data collected in the eCRFs will be captured in a specially constructed and validated database. The data will be validated using both manual and electronic means. Clarification of data will be requested from the Investigator site as required. An audit trail of the original database entries, changes and deletions, session dates and times, and the credentials of the database user who performed the operation will be maintained by the system. The completed database will be quality assured and locked to prevent further changes. A full database extract will be made available for statistical analysis according to the methods outlined in Section 17 and the Statistical Analysis Plan (SAP).

AEs and medical history entries will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO DD). Versions of the dictionaries used will be documented in the Data Management Plan and SAP.

## 17 STATISTICAL METHODS AND PLANNED ANALYSES

This section provides the basis for the SAP for the study. The SAP may be revised during the study to accommodate amendments to the clinical study protocol and to make changes to adapt to unexpected issues in study execution and data that may affect the planned analyses. Any deviations from the planned analysis will be described and justified in a separate document and in the clinical study report (CSR).

The following analyses related to the objectives will be done twice:

Interim Data Lock and Interim Analysis will take place when the 190th subject randomized in Study MT-1186-A02 completes the last visit in that study. At this timepoint, data-lock will combine data collected up to the Week 48 visit in Study MT-1186-A02 with data collected from Study MT-1186-A04. The timing of Study MT-1186-A04 data lock will take place at an appropriate time following completion of the MT-1186-A02 data lock.

The results will not be disclosed to any site-facing personnel or to any personnel directly involved with the conduct of the study.

Final Data Lock and Final Analysis will take place when the last subject completes the Week 50 visit or the safety follow up period of Study MT-1186-A04.

The database locks will be done for each of the above time points, respectively. Each database lock will be associated with a designated SAP that will describe Interim and Final analyses, respectively. Each SAP will be approved and signed prior to the corresponding database lock. Additional analysis may be performed if deemed necessary.

The analysis undertaken for Study MT-1186-A04 will include data from the beginning (baseline) of Study MT-1186-A02 until the end of Study MT-1186-A04. The data will also include information for subjects who early terminated during Study MT-1186-A02 or decided not to continue into Study MT-1186-A04. Further details of which visits in Study MT-1186-A02 will be analyzed for each endpoint will be described in the SAP.

## 17.1 Study Estimands

#### **Primary Estimand**

The primary estimand construction elements are:

- Treatment of interest: The initially randomized treatment Group 1 (edaravone daily) to be compared with Group 2 (edaravone on/off) for up to 96 weeks.
- Population: Subjects with ALS as defined in the analysis set.
- Variable: Time from the randomization date in Study MT-1186-A02 to at least a 12-point decrease in ALSFRS-R or death, whichever happens first.
- Inter-current event (ICE) handling strategy
  - > ICE1 Additional AMX0035 treatment up to 96 weeks double-blind treatment period will be handled using treatment policy strategy.

- ➤ ICE2 Death will be handled within the primary endpoint derivation using composite variable strategy.
- Population-level summary: The Kaplan-Meier estimates and the hazard ratio between Group 1 and Group 2 will be derived from Kaplan-Meier plot and Cox PH regression, respectively.

The treatment effect on the primary endpoint taking death event (ICE2) into account is attributed regardless of the use of additional AMX0035 treatment (ICE1).

## **Secondary Estimand**

The secondary estimand will be tested as supportive analysis for the primary endpoint.

The secondary estimand construction elements are:

- Treatment of interest: as specified for the primary estimand.
- Population: as specified for the primary estimand.
- Variable: as specified for the primary estimand.
- ICE handling strategy
  - > ICE1 Additional AMX0035 treatment up to 96 weeks double-blind treatment period will be handled using hypothetical strategy.
  - > ICE2 Death will be handled within the primary endpoint derivation using composite variable strategy.
- Population-level summary: as specified for the primary estimand.

The above estimand will also be tested when the primary endpoint event is censored if it occurs after ICE1 (additional AMX0035 treatment). In this estimand, the treatment effect will be attributed as if AMX0035 treatment had not been available.

## 17.2 Determination of Sample Size

The sample size for this study is not based on a formal statistical calculation. In total, approximately 300 subjects who have successfully completed Study MT-1186-A02 will be enrolled in this study. However, data from 380 subjects (190 subjects per group) randomized in Study MT-1186-A02 will be included for all analysis. Using Study MT-1186-A02 and MT-1186-A04 survival data, the planned sample size of 190 subjects per group initially randomized in Study MT-1186-A02 will have 70% power to detect a statistically significant result if the true hazard ratio between edaravone 105 mg daily (test) and edaravone 105 mg on/off regimen (control) in the primary endpoint is 0.775, which means 22.5% risk reduction in the hazard due to daily treatment, assuming 65% survival rate at Week 48 for the control group. This calculation of 70% power assumes a 2-sided alpha of 20% based on a rare disease condition, 19 using the log-rank test and a follow-up time of up to 48 weeks in Study MT-1186-A04.

## 17.3 Analysis Sets

The statistical analysis will be based on separate analysis sets, defined as follows:

## Randomized Set:

The randomized set is defined as all of the subjects randomized in Study MT-1186-A02. The subjects will be grouped by the planned treatment allocation (as randomized).

## Efficacy Analysis Set:

The full analysis set (FAS) is defined as all of the subjects randomized in Study MT-1186-A02 who received at least 1 dose of study medication in Study MT-1186-A02 and had any efficacy data collected after randomization. Subjects in the FAS will be grouped and analyzed based on the planned treatment allocated (as randomized). Efficacy endpoints will be analyzed using the FAS.

## Safety Analysis Set:

The Safety Analyses Set (SAF) is defined as all of the subjects randomized in Study MT-1186-A02, and who received at least 1 dose of study drug in Study MT-1186-A02. Subjects will be grouped and analyzed based on the actual treatment received. Safety endpoints will be analyzed using the SAF by treatment group.

## 17.4 Statistical Analyses

#### 17.4.1 General Considerations

The statistical analysis will be performed using SAS® Version 9.4 or higher.

In general, continuous variables will be summarized descriptively using the number of observations (n), mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized using frequency counts and percentages.

Statistical summaries will be presented for the changes from baseline to each visit for the primary, secondary (key and other), and exploratory endpoints that are applicable.

All individual subject data will be listed.

## 17.4.2 Data Handling

## 17.4.2.1 Definition of Baseline for the Efficacy and Safety Endpoints

The data collected before the first study drug dose administration date in Study MT-1186-A02 will be used as the baseline for statistical analysis in Study MT-1186-A04.

## 17.4.2.2 Handling of Time Point Data in Analyses Performed by Measurement Time Point (Analysis Visit Windows)

For the analyses performed for each measurement time point, the allowable range of data handling for the analysis will be specified as analysis visit window in the SAP.

No data imputation will be performed using data from outside the allowable range. If multiple values are available within the allowable range for the endpoint in question, then the latest value will be analyzed.

## 17.4.2.3 Handling of Reference Values and Indeterminate Values for Clinical Laboratory Test Parameters

If a laboratory test value or its reference is indeterminate due to a problem with the test sample, then this value will be handled as a missing value.

## 17.4.3 Statistical Analysis Method

## 17.4.3.1 Subject Disposition

The following will be provided:

- The total number of screened subjects: defined as those who met the inclusion criteria regarding the target indication and signed the ICF
- The total number of subjects enrolled
- The total number (%) of subjects in each analysis set
- The total number (%) of subjects who completed Week 48
- The total number (%) of subjects who discontinued the study, and the reasons for discontinuation

## 17.4.3.2 Concomitant Medications

All concomitant medications will be coded using the WHO DD and anatomical therapeutic chemical (ATC) system. Concomitant medication is defined as any medication, other than study drug, which is taken after the first dose administration in Study MT-1186-A02. Concomitant medications, except for riluzole, will be summarized by ATC level 2 categories and preferred name.

Riluzole and AMX0035 administration will be summarized separately.

## 17.4.4 Study Medication Exposure

The duration of exposure in days will be calculated as follows:

Date of last dose of edaravone in Study MT-1186-A04 – date of first dose of edaravone in Study MT-1186-A02 + 1

If the date of first dose or the date of last dose cannot be determined, the duration calculation will not be completed. The duration of exposure will be summarized using descriptive statistics.

All exposure data will be listed. Interruptions and compliance are not considered for the duration of exposure.

## 17.4.5 Efficacy Analysis

## 17.4.5.1 Primary Efficacy Analysis

Data of time from randomization in Study MT-1186-A02 to at least a 12-point decrease in ALSFRS-R or death will be included regardless of AMX0035 use (ICE1). In other words, data following AMX0035 treatment will be used in the analysis and will not be censored.

The primary efficacy endpoints associated with the study estimand will be analyzed on the randomized set using Kaplan-Meier estimates, 2-sided alpha with a nominal 20% significance level and 80% CIs. The comparison between Treatment Group 2 versus Treatment Group 1 will be performed using a log rank test with Study MT-1186-A02 randomization strata of ALSFRS-R rate of decline score from the MT-1186-A02 screening period (2 levels strata of -1,-2 or -3,-4) and the geographical region (3 levels strata of Europe, America, or Asia Pacific). Subjects without events during treatment will be right censored at the date of last study visit.

## 17.4.5.2 Supportive Analyses for the Primary Efficacy Endpoint

The primary efficacy endpoint will also be analyzed using the Cox Proportional Hazard (COX PH) Model with terms for treatment as explanatory variable and baseline ALSFRS-R score, and the MT-1186-A02 randomization strata as covariates. This statistical test will be done as 2-sided with a nominal 20% significance level. Point estimates of treatment differences will be accompanied with 2-sided 80% CIs.

## 17.4.5.3 Supportive Analysis for the Secondary Estimand

The primary analysis will be repeated when the event of interest is censored if it occurs after initiation of AMX0035 treatment, using the Inverse Probability of Censoring Weighting (IPCW by Robins JM, Finkelstein et all, 2000)<sup>20</sup> to adjust for non-random time-dependent covariates. Further details on this supportive analysis will be specified in the Statistical Analysis Plan.

## 17.4.5.4 Efficacy Analyses for Secondary Endpoints

CAFS analysis ranks clinical outcomes on the basis of survival time and change in the ALSFRS-R score will be analyzed at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04. In this analysis, a subject's score will be calculated by comparing each subject to every other subject within each treatment group in the study, resulting in a score of +1 if the outcome was better than the subject being compared, -1 if worse, and 0 if the same. The subject's score will then be calculated by summing up their comparison to all of the other subjects within each treatment group in the study as CAFS score. A subject who dies earlier than the comparator subject will be given a comparison score of -1. For a subject who discontinues early for a reason other than death, that subject and the comparator's score will be based on the change from baseline of the ALSFRS-R score at the latest timepoint at which they both have an ALSFRS-R score. In general, these comparisons will result in subjects who die being assigned the worst scores and ranked according to the time of death. Subjects who survive and complete the study will be ranked more favorably than subjects who die. The CAFS score will be evaluated at all visits from

baseline in Study MT-1186-A02 to the end of Study MT-1186-A04 using an ANCOVA model with treatment group and Study MT-1186-A02 randomization strata as fixed effects, and baseline ALSFRS-R total score as covariate. The difference between the 2 treatment groups in the CAFS scores will be also compared using the generalized Gehan-Wilcoxon test as a sensitivity analysis.

The following sequence of parametric and semi-parametric models will be conducted to estimate the clinical benefit:

- Mixed-effect model for repeated measure (MMRM) as specified below.
- COX PH model as specified above.

Change in ALSFRS-R score will be analyzed at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04 using MMRM with terms for baseline ALSFRS-R score, Study MT-1186-A02 randomization strata, treatment, visit, and treatment-by-visit interaction. The unstructured covariance matrix will be used to model the within-subject errors. Denominator degrees of freedom will be estimated using Kenward-Roger's approximation. The least-squares mean estimates for the mean change at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04, as well as the difference of the estimates between oral edaravone 105 mg daily versus oral edaravone 105 mg on/off regimen, will be displayed with their corresponding standard errors, p-values, and 95% CI.

## 17.4.5.5 Efficacy Analyses for Other Secondary Exploratory Endpoints

The following endpoints with continuous values will be analyzed using the same method (MMRM) and the same survival analysis as specified above:

- 1. Time from the randomization date in Study MT-1186-A02 to death, tracheostomy, or permanent assisted mechanical ventilation (≥23 hours/day)
- 2. Change in %SVC at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04
- 3. Change in body weight at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04
- 4. Time from the randomization date in Study MT-1186-A02 to death or permanent assisted mechanical ventilation (≥23 hours/day)
- 5. Time from the randomization date in Study MT-1186-A02 to death
- 6. Change in ALSAQ40 at all visits from baseline in Study MT-1186-A02 to the end of Study MT-1186-A04

## 17.4.5.6 Efficacy Analyses for Other Exploratory Endpoints

King's ALS Clinical Stage will be derived from ALSFRS-R score and death. The frequency and percent for King's ALS Clinical Stage at each visit will be provided by each treatment group using shift tables.

## 17.4.5.7 Type I Error Control

Since no formal hypothesis was formulated, type I error will not be controlled. Unless otherwise specified, all statistical tests for the primary endpoint and the other endpoints will be done as 2-sided with a nominal 20% and 5% significance level, respectively. Point estimates of treatment differences will be accompanied with 2-sided 80% and 95% confidence intervals where applicable, respectively.

## 17.4.5.8 Safety Analyses

An AE will be considered a TEAE if:

- 1) The AE was not present before the first dose in Study MT-1186-A02 but started after administration of the first dose of study drug in Study MT-1186-A02, or
- 2) The AE was present before the first dose in Study MT-1186-A02 but increased in severity following administration of the first dose of study drug in Study MT-1186-A02.

TEAEs will be coded using the latest available version of MedDRA and will be summarized in incidence tables by System Organ Class (SOC) and Preferred Term (PT). The numbers and proportions of subjects with TEAEs will be calculated for each treatment group by SOC and PT.

The following summaries will be presented:

- TEAEs by SOC and PT
- TEAEs by SOC, PT, and severity
- TEAEs by SOC, PT, and drug relationship
- TEAEs leading to discontinuation of study drug by SOC and PT
- TEAEs leading to death by SOC and PT
- TEAEs related to study drug by SOC, PT, and severity
- TEAEs of Peripheral Neuropathy Standardized MedDRA query by SOC and PT
- Serious TEAEs by SOC and PT
- Serious TEAEs related to study drug by SOC and PT

For each of the summaries, multiple occurrences of the same event within a subject will be counted once in the summaries by SOC and PT; multiple occurrences of the same event within a subject will be counted once in the maximum severity category (severe>moderate>mild) and/or maximum study drug relationship category (reasonable possibility/no reasonable possibility). If severity or relationship is found to be missing, the most severe occurrence will be imputed for that summary.

All AEs for each subject, including multiple occurrences of the same event, will be presented in full in a comprehensive listing including subject number, severity, seriousness, action taken, outcome, relationship to treatment, onset/stop date, and duration.

Duration of the AE and time to the AE occurrence from start of edaravone will be calculated and presented in days (duration = AE stop date - AE start date + 1 and time to AE occurrence = AE start date - The first administration date of study drug + 1).

## 17.4.5.9 Other Safety Analyses

## 12-lead ECG

The 12-lead ECG parameters (RR interval, heart rate, QRS, QT, QTcB, and QTcF) will be descriptively summarized for values and changes from baseline.

For evaluation ("Normal/abnormal CS/abnormal NCS") by the Investigator of 12-lead ECG, the number and percentage of subjects with each category will be summarized at each visit.

## **Vital Signs**

Vital signs (sitting systolic and diastolic blood pressure, heart rate, respiratory rate, and axillary, oral, temporal [skin-based], or tympanic body temperature) will be descriptively summarized for values and changes from baseline at each visit.

For evaluation ("Normal/abnormal CS/abnormal NCS") of vital signs by the Investigator, a shift table of the change from baseline will be summarized at each visit by treatment group.

## **Clinical Laboratory Assessments**

Clinical laboratory tests described in Section 13.5 will be descriptively summarized for values and the changes from baseline at each visit by each treatment group. For urinalysis parameters, shift tables will be prepared for each visit and category by treatment group.

#### C-SSRS

For the C-SSRS, the number and percentage of subjects with suicidal ideation or suicidal behavior as recorded on the C-SSRS scale will be presented by treatment group. The distribution of responses for most severe suicidal ideation and suicidal behavior during the treatment period will be summarized by treatment group.

# 18 STUDY MANAGEMENT AND ETHICAL AND REGULATORY REQUIREMENTS

## 18.1 Good Clinical Practice

The Investigator will ensure that this study is conducted in compliance with the 2013 (Fortaleza, Brazil) revision of the 1964 Declaration of Helsinki. This study will also be conducted in accordance with GCP requirements described in the current revision of ICH of Technical Requirements of Pharmaceuticals for Human Use Guidelines. This study will also be carried out in accordance with regional and local legal requirements. Before the first subject is enrolled in the study, all ethical and legal requirements will be met.

## 18.2 Investigator Responsibilities

#### 18.2.1 Informed Consent Form

Prior to undergoing any study-specific procedure, all subjects or their LAR must consent in writing to participate. An ICF will be given to each subject, which will contain all regulatory-required elements, all ICH-required elements, and data protection information, when applicable, in a language that is understandable to the subject or their LAR.

The process of obtaining the ICF will follow all regulatory regulations, ICH requirements, and local laws.

Either the Investigator or a designated person, qualified to meet any applicable local regulations and who is equally knowledgeable about the study, will explain the aims, methods, anticipated benefits and potential hazards of the study and any discomfort it may entail. The review must be in a form understandable to the subject or their LAR. A corresponding written explanation will also be provided, and the subject allowed sufficient time to consider the study information.

If the subject is willing to participate in the study, the ICF will be signed and dated by the subject, the Investigator or, if applicable, the designated person who explained the nature of the study. The subject will receive a copy (together with the information sheet) and the original ICF will be retained with the study records at the Investigator site.

If the subject is unable to personally sign and write their name and date on the ICF because ALS is affecting their ability to write, the subject's LAR can sign and date the form on behalf of the subject. The LAR must verify that the subject has heard and was provided with all of the necessary information and that all of their questions were answered satisfactorily by the Investigator, after which the subject voluntarily gave their consent by some other means (e.g., speaking, nodding, blinking).

The date (and time, if required) on which the ICF is signed by the subject must be recorded in the source notes.

The Investigator or his/her designee must emphasize to the subject that study participation is entirely voluntary and that consent regarding study participation may be withdrawn at any time without penalty or loss of benefits to which the subject is otherwise entitled.

If the ICF is amended during the study, the Investigator must follow all applicable regulatory requirements pertaining to approval of the amended ICF by the IRB/IEC. The Investigator site personnel must use the amended ICF for all new subjects and repeat the consent process with the amended ICF for any ongoing subjects.

## 18.2.2 Ethical and Regulatory Approval

The study will be conducted in accordance with ethical principles that have their origins in the Declaration of Helsinki and that are consistent with GCP as described in:

- 1. Declaration of Helsinki, concerning medical research in humans (Adopted by the 18th World Medical Association [WMA] General Assembly, Helsinki, Finland, June 1964 and amended by the: 29th WMA General Assembly, Tokyo, Japan, October 1975; 35th WMA General Assembly, Venice, Italy, October 1983; 41st WMA General Assembly, Hong Kong, September 1989; 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996; 52nd WMA General Assembly, Edinburgh, Scotland, October 2000; 53rd WMA General Assembly, Washington DC, USA, October 2002 (Note of Clarification added); 55th WMA General Assembly, Tokyo, Japan, October 2004 (Note of Clarification added); 59th WMA General Assembly, Seoul, Republic of Korea, October 2008; 64th WMA General Assembly, Fortaleza, Brazil, October 2013).
- 2. ICHE6 R2
- 3. Directive 91/507/European Economic Community, The Rules Governing Medicinal Products in the European Community
- 4. The Medicines for Human Use (Clinical Trials) Regulations 2004 (Statutory Instrument 2004 No 1031) and subsequent amendments
- 5. Association of the British Pharmaceutical Industry Guidelines for Phase 1 Trials (2012)
- 6. EMEA, Committee for Medicinal Products for Human Use (CHMP). September 2007. Guideline on Strategies to Identify and Mitigate Risks for First-in-Human Clinical Trials with IMPs. (EMEA/CHMP/Safety Working Party/28367/07).
- 7. CFR Title 21

The Investigator and Sponsor will sign this Protocol to confirm agreement to abide by it. A Coordinating Investigator will be identified and appointed to sign the CSR.

Before any study-related procedure is performed on a subject, all IRB/IEC, regulatory and local approvals of this Protocol will be obtained. While the study is ongoing and at study completion/discontinuation, the Sponsor or Investigator will submit information to the IRB/IEC(s) in accordance with institutional/local regulations, for example:

- Information on SUSARs
- Periodic reports on the progress of the study
- Notification of the EOS or ET
- Final study summary upon completion or closure.

The Sponsor will ensure that any SUSARs from this study and other studies with this IMP are reported promptly to the regulatory authorities.

If it is necessary to amend the Protocol during the study, proper notification will be made to the regulatory authorities and IRB/IECs in the form of a Protocol Modification. Protocol
Modification requiring IRB/IEC approval may be implemented only after a copy of the IRB/IEC's approval/favorable opinion letter has been transmitted to the Sponsor and regulatory authority approval has been obtained (if required). Protocol Modifications that are intended to eliminate an apparent immediate hazard to subjects may be implemented prior to receiving Sponsor, regulatory authority and/or IRB/IEC approval. However, in this case, approval must be obtained as soon as possible after implementation.

Any Protocol or other deviations that occur during the study will be documented and reported to the Sponsor. Depending on the nature of the deviation, this may be reported to the appropriate regulatory authority and IRB/IEC.

#### 18.2.3 Source Document Requirements and Document Access During the Study

The Investigator must retain a comprehensive and centralized filing system of all study-related documentation (including, but not limited to: essential documents, copies of Protocols, eCRFs, source data such as original reports of test results, IMP dispensing logs, correspondence, records of ICF and other documents pertaining to the conduct of the study) that is suitable for inspection by the Sponsor and representatives of regulatory authorities.

The Investigator/institution will permit study-related monitoring, audits, IRB/IEC reviews, and regulatory inspections providing direct access to source data/documents.

#### 18.2.4 Study Records Retention

Study-related documentation must be kept for at least 25 years or until notified by the Sponsor. Documents should be stored in such a way that they can be accessed/data retrieved at a later date. Consideration should be given to security and environmental risks.

No study document will be destroyed without prior written agreement between the Sponsor and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, written agreement must be obtained from the Sponsor.

#### 18.3 Study Monitoring

In accordance with applicable regulations, GCP and the procedures of the Sponsor or its designees, the Study Monitor will periodically contact the Investigator site, and conduct on-site visits. The extent, nature and frequency of on-site visits will be based on study complexity, enrollment rate and data quality at the Investigator site. Through these visits and frequent communications (e.g., letter, email, and telephone), the Study Monitor will verify that the study is conducted according to Protocol, regulatory and Sponsor requirements.

The Investigator will allow the Study Monitor direct access to all relevant documents and allocate his/her time and the time of his/her personnel to the Study Monitor to discuss findings and any relevant issues.

In addition to contacts during the study, the Study Monitor will contact the Investigator site personnel prior to the start of the study to discuss the Protocol and data collection procedures.

At study closure, the Study Monitor will conduct all activities as indicated in Section 18.5.

#### 18.4 Quality Assurance and Auditing

Authorized representatives of the Sponsor, IRB/IEC and/or regulatory authorities may conduct an audit or inspection of this study either during or after completion. In such cases, the Investigator will give the auditor/inspector direct access to all relevant documents and source data and will allocate his/her time and the time of his/her personnel as may be required to discuss findings and any relevant issues.

#### 18.5 End-of-study and Site Closure

The end of the study is defined as the last visit for the last subject. Upon completion of the study, or if the study or an Investigator site is prematurely discontinued, the following activities, where applicable, must be conducted by the Study Monitor in conjunction with the Investigator:

- Return of all study data to the Sponsor
- Completion of data clarifications and/or resolutions
- Accounting, reconciliation, and final disposition of used and unused IMP
- Review of Investigator site study records for completeness

Any unresolved AEs or SAEs will be followed according to Section 15.8.

#### 18.6 Premature Discontinuation of the Study

The Sponsor reserves the right to discontinue the study because of safety concerns, ethical issues, or serious and/or persistent non-compliance with the Protocol.

If the study is suspended or terminated, the Sponsor will promptly inform the Investigator, and will also inform the regulatory authorities of the suspension or termination of the study and the reason(s) for the action. The Investigator is responsible for promptly informing the IRB/IEC and providing the reason(s) for the suspension or termination of the study.

For all subjects, the Follow-up visit assessments should be performed per Table 1.

In addition, all general Investigator site activities required for the scheduled EOS and site closure should be completed, as described in Section 18.5.

The Sponsor may at any time, at its sole discretion, discontinue the study for various reasons, including, without limitation, the following:

- Failure of the Investigator to enroll subjects into the study at a reasonable rate
- Failure of the Investigator to comply with applicable laws and/or pertinent regulations
- Submission of knowingly false information from the research facility to the Sponsor, Study Monitor, or regulatory authorities
- Insufficient adherence to Protocol requirements.

The Sponsor will issue a written notice to the Investigator, which will contain the reasons for taking such action. If the Investigator site is terminated for non-compliance, appropriate regulatory authorities will also be notified by the Sponsor.

### 18.7 Liability and Insurance

Refer to the written study information given to the subject.

#### 19 DISCLOSURE OF DATA

#### 19.1 Confidentiality

A Subject Screening and Enrollment Log will be completed at each Investigator site for all subjects who signed an ICF. A Subject Identification Log, documenting the subjects' names, will be completed, and retained at each Investigator site for all subjects enrolled in the study.

Subject names will remain confidential and will not be included in the database supplied to the Sponsor or its designee. If the subject name appears on any document collected, e.g., hospital discharge summary, the name must be redacted before the document is transmitted to the Sponsor or its designee. All study findings will be stored in electronic databases. The subjects will give explicit permission for representatives of the Sponsor, regulatory authorities, and the IRB/IEC to inspect their medical records to verify the information collected. Subjects will be informed that all personal information made available for inspection will be handled in the strictest confidence and in accordance with laws and regulations. All personnel involved in the study will observe and work within the confines of local data protection regulations.

All information concerning the product as well as any information such as clinical indications for the IMP, its formula, methods of manufacture and other scientific data relating to it, that have been provided by the Sponsor or designee, are confidential and are the sole property of the Sponsor. The Investigator will agree to use the information only for the purposes of carrying out this study and for no other purpose unless prior written permission from the Sponsor is obtained. The Sponsor has full ownership of the eCRFs completed as part of the study.

#### 19.2 Publication

By signing the study Protocol, the Investigator agrees that the results of the study may be used for the purposes of national registration, publication, and information for medical and pharmaceutical professionals by the Sponsor. If necessary, the regulatory authorities will be notified of the Investigator's name, address, qualifications, and extent of involvement.

The Sponsor will retain ownership of all data. All proposed publications based on the study will be subject to the Sponsor's approval requirements.

The Sponsor or designee will prepare a final report on the study. The Investigator's right to publish or present any information on the study, and publication procedures to be followed, will be defined in the Investigator site agreement.

#### 20 LIST OF REFERENCES

- 1. Traynor B, Alexander M, Corr B, Frost E, Hardiman O. Effect of a multidisciplinary amyotrophic lateral sclerosis (ALS) clinic on ALS survival: a population based study, 1996–2000. Journal of Neurology, Neurosurgery & Psychiatry. 2003;74(9):1258-61.
- 2. Miller RG, Jackson CE, Kasarskis EJ, England JD, Forshew D, Johnston W, et al. Practice parameter update: the care of the subject with amyotrophic lateral sclerosis: drug, nutritional, and respiratory therapies (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2009;73(15):1218-26.
- 3. Miller RG, Jackson CE, Kasarskis EJ, England JD, Forshew D, Johnston W, et al. Practice Parameter update: the care of the subject with amyotrophic lateral sclerosis: multidisciplinary care, symptom management, and cognitive/behavioral impairment (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2009;73(15):1227-33.
- 4. EFNS Task Force on Diagnosis, Management of Amyotrophic Lateral S, Andersen PM, Abrahams S, Borasio GD, de Carvalho M, et al. EFNS guidelines on the clinical management of amyotrophic lateral sclerosis (MALS)--revised report of an EFNS task force. Eur J Neurol. 2012;19(3):360-75.
- 5. Brooks BR. El Escorial World Federation of Neurology criteria for the diagnosis of amyotrophic lateral sclerosis. Subcommittee on Motor Neuron Diseases/Amyotrophic Lateral Sclerosis of the World Federation of Neurology Research Group on Neuromuscular Diseases and the El Escorial "Clinical limits of amyotrophic lateral sclerosis" workshop contributors. J Neurol Sci. 1994;124 Suppl:96-107.
- 6. Brooks BR, Miller RG, Swash M, Munsat TL, World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000;1(5):293-9.
- 7. Millul A, Beghi E, Logroscino G, Micheli A, Vitelli E, Zardi A. Survival of subjects with amyotrophic lateral sclerosis in a population-based registry. Neuroepidemiology. 2005;25(3):114-9.
- 8. Qureshi M, Schoenfeld DA, Paliwal Y, Shui A, Cudkowicz ME. The natural history of ALS is changing: improved survival. Amyotrophic Lateral Sclerosis. 2009;10(5-6):324-31.
- 9. Abe K, Itoyama Y, Sobue G, Tsuji S, Aoki M, Doyu M, et al. Confirmatory double-blind, parallel-group, placebo-controlled study of efficacy and safety of edaravone (MCI-186) in amyotrophic lateral sclerosis subjects. Amyotroph Lateral Scler Frontotemporal Degener. 2014;15(7-8):610-7.
- 10. Edaravone ALS 16 Study Group. A post-hoc subgroup analysis of outcomes in the first phase III clinical study of MT-1186 (MCI-186) in amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2017;18(sup1):11-9.
- 11. Writing Group on behalf of the edaravone (MCI-186) ALS 19 Study Group. Safety and efficacy of edaravone in well-defined subjects with amyotrophic lateral sclerosis: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2017;16(7):505-12.
- 12. Writing Group on behalf of the edaravone ALS 17 Study Group. Exploratory double-blind, parallel-group, placebo-controlled extension study of edaravone

- (MCI-186) in amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2017;18(sup1):20-31.
- Writing Group on behalf of the edaravone ALS 19 Study Group. Open-label 24-week extension study of edaravone (MCI-186) in amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2017;18(sup1):55-63.
- 14. Takei K, Watanabe K, Yuki S, Akimoto M, Sakata T, Palumbo J. Edaravone and its clinical development for amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2017;18(sup1):5-10.
- 15. US Food and Drug Administration (FDA). Center for Drug Evaluation and Research. Application number: 209176Orig1s000: Clinical Pharmacology and Biopharmaceutics Review(s). 2017.
- 16. Edaravone Investigator Brochure, June 2022 version 4.
- 17. Quanjer P, Stanojevic S, Cole T, Baur X, Hall G, Culver B, et al, Multi-ethnic reference values for spirometry for the 3-95 year age range: the global lung function 2012 equations: Report of the Global Lung Function Initiative (GLI), ERS Task Force to established improved Lung Function Reference Values. Eur Respir J. 2012;40(6):1324-1343.
- 18. Blendra R, Leigh N, Jackson C, et al, Estimating clinical stage of amyotrophic lateral sclerosis from ALS Functional Rating Scale. Amyotroph Lateral Scler Frontotemporal Degener. 2014;15 (3-4):279-284.
- 19. Hilgers RD, Roes K, Stallard N, IDeAI, Asterix and InSPiRe project groups. Directions for new developments on statistical design and analysis of small population group trials. Orphanet J Rare Dis. 2016;11(1):78.
- 20. Robins JM, Finkelstein DM. Correcting for non-compliance and dependent censoring in an AIDS Clinical Trial with inverse probability of censoring weighted (IPCW) log-rank tests. Biometrics 2000;56:779-788.

#### 21 APPENDICES

## APPENDIX 1 EL ESCORIAL REVISED CRITERIA FOR DIAGNOSIS OF AMYOTROPHIC LATERAL SCLEROSIS (EXAMPLE)

#### The diagnosis of amyotrophic lateral sclerosis (ALS) requires:

#### A - the presence of:

- (A:1) evidence of *lower motor neuron degeneration (LMN)* by clinical, electrophysiological or neuropathologic examination,
- (A:2) evidence of upper motor neuron degeneration (UMN) by clinical examination, and
- (A:3) progressive spread of symptoms or signs within a region or to other regions, as
- determined by history or examination,

#### together with B - the absence of:

- (B:1) electrophysiological and pathological evidence of other disease processes that might explain the signs of LMN and/or UMN degeneration, and
- (B:2) neuroimaging evidence of other disease processes that might explain the observed clinical and electrophysiological signs.

A careful history, physical and neurological examination must search for clinical evidence of UMN and LMN signs in 4 regions of the central nervous system: brainstem, cervical, thoracic, or lumbosacral spinal cord (see Table below). Ancillary tests should be reasonably applied, as clinically indicated, to exclude other disease processes. These should include electro diagnostic, neurophysiological, neuroimaging and clinical laboratory studies.

Lower Motor Neuron and Upper Motor Neuron Signs in Four Central Nervous System Regions

| | Brainstem | Cervical | Thoracic | Lumbosacral |
|---|---|---|---|---|
| Lower motor<br>neuron signs<br>weakness, atrophy,<br>fasciculations | Jaw, face, palate, tongue, larynx | neck, arm, hand,<br>diaphragm | back,<br>abdomen | back, abdomen, leg,<br>foot |
| Upper motor neuron signs, pathologic spread of reflexes, clonus, etc. | Clonic jaw, gag reflex,<br>exaggerated snout reflex,<br>pseudobulbar features,<br>forced yawning,<br>pathologic DTRs, spastic<br>tone | Clonic DTRs,<br>Hoffman reflex,<br>pathologic DTRs,<br>spastic tone,<br>preserved reflex in<br>weak wasted limb | Loss of superficial abdominal reflexes, pathologic DTRs, spastic tone | Clonic DTRs -extensor<br>plantar response,<br>pathologic DTRs, spastic<br>tone, preserved reflex in<br>weak wasted limb |

Abbreviation: DTR=deep tendon stretch reflex

#### Clinical evidence of LMN and UMN degeneration is required for the diagnosis of ALS.

The clinical diagnosis of ALS, without pathological confirmation, may be categorized into various levels of certainty by clinical assessment alone depending on the presence of UMN and LMN signs together in the same topographical anatomic region in either the brainstem (bulbar cranial motor neurons), cervical, thoracic, or lumbosacral spinal cord (anterior horn

Confidential

motor neurons). The terms Clinical Definite ALS and Clinically Probable ALS are used to describe these categories of clinical diagnostic certainty on clinical criteria alone:

Clinically Definite ALS is defined on clinical evidence alone by the presence of UMN, as well as LMN signs, in 3 regions.

Clinically Probable ALS is defined on clinical evidence alone by UMN and LMN signs in at least 2 regions with some UMN signs necessarily rostral to (above) the LMN signs.

Clinically Probable - Laboratory-Supported ALS is defined when clinical signs of UMN and LMN dysfunction are in only 1 region, or when UMN signs alone are present in 1 region, and LMN signs defined by electromyography criteria are present in at least 2 limbs, with proper application of neuroimaging and clinical laboratory protocols to exclude other causes.

Clinically Possible ALS is defined when clinical signs of UMN and LMN dysfunction are found together in only 1 region or UMN signs are found alone in 2 or more regions; or LMN signs are found rostral to UMN signs and the diagnosis of Clinically Probable – Laboratory supported ALS cannot be proven by evidence on clinical grounds in conjunction with electro diagnostic, neurophysiologic, neuroimaging or clinical laboratory studies. Other diagnoses must have been excluded to accept a diagnosis of clinically possible ALS.

Clinically Suspected ALS it is a pure LMN syndrome, wherein the diagnosis of ALS could not be regarded as sufficiently certain to include the subject in a research study. Hence, this category is deleted from the revised El Escorial Criteria for the Diagnosis of ALS.

## APPENDIX 2 ALS FUNCTIONAL RATING SCALE- REVISED (ALSFRS-R) (EXAMPLE)

| 1 Speech | 6 Dressing and hygiene |
|---|---|
| 4: Normal speech processes | 4: Normal function |
| 3: Detectable speech disturbance | 3: Independent and complete self-care with effort or decreased efficiency |
| 2: Intelligible with repeating | 2: Intermittent assistance or substitute methods |
| 1: Speech combined with nonvocal communication | 1: Needs attendant for self-care |
| 0: Loss of useful speech | 0: Total dependence |
| 2 Salivation | 7 Turning in bed and adjusting bed clothes |
| 4: Normal | 4: Normal |
| 3: Slight but definite excess of saliva in mouth; may have nighttime drooling | 3: Somewhat slow and clumsy, but no help needed |
| 2: Moderately excessive saliva; may have minimal drooling | 2: Can turn alone or adjust sheets, but with great difficulty |
| 1: Marked excess of saliva with some drooling | 1: Can initiate, but not turn or adjust sheets alone |
| 0: Marked drooling; requires constant tissue or handkerchief | 0: Helpless |
| 3 Swallowing | 8 Walking |
| 4: Normal eating habits | 4: Normal |
| 3: Early eating problems — occasional choking | 3: Early ambulation difficulties |
| 2: Dietary consistency changes | 2: Walks with assistance |
| 1: Needs supplemental tube feeding | 1: Nonambulatory functional movement |
| 0: NPO (exclusively parenteral or enteral feeding) | 0: No purposeful leg movement |
| 4 Handwriting | 9 Climbing stairs |
| 4: Normal | 4: Normal |
| 3: Slow or sloppy: all words are legible | 3: Slow |
| 2: Not all words are legible | 2: Mild unsteadiness or fatigue |
| 1: Able to grip pen but unable to write | 1: Needs assistance |
| 0: Unable to grip pen | 0: Cannot do |
| 5a Cutting food and handling utensils (subjects without gastrostomy)? | 10 Dyspnea |
| 4: Normal | 4: None |
| 3: Somewhat slow and clumsy, but no help needed | 3: Occurs when walking |
| 2: Can cut most foods, although clumsy and slow; some help needed | 2: Occurs with 1 or more of the following: eating, bathing, dressing (ADL) |
| 1: Food must be cut by someone, but can still feed slowly | 1: Occurs at rest, difficulty breathing when either sitting or lying |
| 0: Needs to be fed | 0: Significant difficulty, considering using mechanical respiratory support |
| 5b Cutting food and handling utensils | 11 Orthopnea |

#### Protocol MT-1186-A04

| (alternate scale for subjects with gastrostomy)? | |
|---|---|
| 4: Normal | 4: None |
| 3: Clumsy but able to perform all manipulations independently | 3: Some difficulty sleeping at night due to shortness of breath, does not routinely use more than 2 pillows |
| 2: Some help needed with closures and fasteners | 2: Needs extra pillows in order to sleep (more than 2) |
| 1: Provides minimal assistance to caregiver | 1: Can only sleep sitting up |
| 0: Unable to perform any aspect of task | 0: Unable to sleep |
| | 12 Respiratory insufficiency |
| | 4: None |
| | 3: Intermittent use of BiPAP |
| | 2: Continuous use of BiPAP during the night |
| | 1: Continuous use of BiPAP during the night and day |
| | 0: Invasive mechanical ventilation by intubation or tracheostomy |

Abbreviations: ADL = activities of daily living; BiPAP = Bi-level Positive Airway Pressure

#### APPENDIX 3 SUBJECT CONTRACEPTION

#### Contraception

Female subjects of child-bearing potential\* must be willing and able to practice birth control for the duration of the study, from the Day 1/screening visit until 3 months after the last dose of IMP. Male subjects must be willing and able to practice birth control for the duration of the study, from the Day 1/screening visit until 3 months after the last dose of IMP.

- Female subjects must be willing to use a highly effective method of birth control (i.e., contraceptive measure with a failure rate of <1% per year), in conjunction with male barrier contraception (i.e., male condom with spermicide). Highly effective methods of contraception include:
  - o Placement of an intrauterine device or intrauterine system.
  - o Established use of oral, injected, or implanted hormonal methods of contraception associated with inhibition of ovulation.
  - o Male sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). (For female subjects on the study, the vasectomized male partner should be the sole partner for that subject.)
  - o Bilateral tubal ligation.
  - O True abstinence: when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

Females must not donate ova for the duration of the study, from the time of the first dose of IMP until 3 months after the last dose of IMP.

- Male subjects with partners of child-bearing potential must use a barrier method of
  contraception (i.e., male condom with spermicide) in addition to a second method of
  acceptable contraception used by their female partners. In addition to the list of highly
  effective contraception methods above, other acceptable methods of contraception
  include:
  - o Progesterone only oral contraception, where inhibition of ovulation is not the primary mode of action.
  - o Cap, diaphragm, or sponge with spermicide.

Male subjects must not donate sperm for the duration of the study, from the time of the first dose of IMP until 3 months after the last dose of IMP.

- \*Note: Women are considered to be of child-bearing potential unless they meet one of the following criteria as documented by the Investigator:
- Post-menopausal for at least 1 year.
- Hysterectomy, bilateral oophorectomy, or salpingectomy.
- Congenital sterility.

Subjects must not have unprotected sexual intercourse with a female who is pregnant or breastfeeding during the study.

## APPENDIX 4 AMYOTROPHIC LATERAL SCLEROSIS ASSESSMENT QUESTIONNAIRE (ALSAQ) 40 (EXAMPLE)

## THE ALS ASSESSMENT QUESTIONNAIRE (ALSAQ 40)

- Please complete this questionnaire as soon as possible. If you have any difficulties filling in the questionnaire by yourself, please get someone else to help you with it. However it is your responses that we are interested in.
- The questionnaire consists of a number of statements about difficulties that you may have experienced during the last 2 weeks. There are no right or wrong answers, your first response is likely to be the most accurate for you. Please tick the box which best describes your own experience or feelings.
- Please try to answer every question even though some may seem rather similar to others, or may not seem relevant to
  you.
- All the information you give will be treated in the strictest confidence, and is completely anonymous. There is no way
  of identifying you from the questionnaire.

The following statements all refer to difficulties that you may have had walking during the last 2 weeks. Please indicate, by ticking the appropriate box, how often the following statements have been true for you.

If you are not able to walk at all please tick Always/cannot walk at all. How often during the last 2 weeks Please tick one box for each question have the following been true? Always/ Sometimes Often Cannot walk Never Rarely at all 1. I have found it difficult to walk short distances, e.g. around the 2. I have fallen over whilst walking. 3. I have stumbled or tripped whilst walking. 4. I have lost my balance whilst walking. 5. I have had to concentrate whilst walking. 6. Walking has tired me out. 7. I have had pains in my legs whilst walking.

Please check that you have ticked one box for each question before going on to the next page

The following statements all refer to certain difficulties that you may have had during the last 2 weeks. Please indicate, by ticking the appropriate box, how often the following statements have been true for you. If you cannot do the activity at all please tick Always/cannot do at all. ~ How often during the last 2 weeks have the following been true? Please tick one box for each question Always/ Never Sometimes Often Cannot do at all 8. I have found it difficult to go up and down the stairs. 9. I have found it difficult to stand up. 10. I have found it difficult to get myself up out of chairs. 11. I have had difficulty using my arms and hands. 12. I have found turning and moving in bed difficult. 13. I have found picking things up difficult. 14. I have found holding books or newspapers, or turning pages difficult. 15. I have had difficulty writing clearly. 16. I have found it difficult to do jobs around the house. 17. I have found it difficult to feed myself.

> Please check that you have ticked <u>one box for each question</u> before going on to the next page

 I have had difficulty combing my hair or cleaning my teeth.

| | If you cannot do the a | ctivity at all pi | ease tick <b>Always</b> /c | cannot do at | all |
|---|---|---|---|---|---|
| low often during the last 2 weeks<br>are the following been true? | | Please tick one box for each question | | | |
| | Never | Rarely | Sometimes | Often | Always/<br>Cannot do<br>at all |
| I have had difficulty getting dressed. | | | | | |
| 1 have had difficulty washing<br>at the hand basin. | | | | | |
| I have had difficulty swallowing. | | | | | |
| 2. I have had difficulty cating solid food. | | | | | |
| 23. I have found it difficult to drink liquids. | | | | | |
| the following statements all refer to cate, by ticking the appropriate box, h | ertain difficulties t<br>ow often the follow | hat you may<br>dog statemer | its have been tru | e tor you. | weeks, Please |
| | Never | Please tie<br>Rarely | k one box for each<br>Sometimes | Often | Always |
| nave the following been true? | Never | | | Often | Always |
| awe the following been true? 24. I have found it difficult to participate in conversations. | Never | | | Often | Always |
| 25. I have felt that my speech has | Never | | | Often | Always |

Please check that you have ticked <u>one box for each question</u> before going on to the next page

| | Never | Rarely | Sometimes | Often | Always |
|---|---|---|---|---|---|
| 28. I have talked less than I used to. | <u> </u> | | | | [] |
| | T. | | | 2 BAAR 2 74 78 | |
| 29. I have been frustrated by my | | | - | | |
| speech. | | | | | |
| 30. I have felt self-conscious about | | | | | |
| my speech. | | | | | |
| | | | <u> </u> | | |
| 31. I have felt lonely. | | | | | |
| | | | p | | |
| 32. I have been bored. | | | | | |
| 33. I have felt embarrassed in | | | | | |
| social situations. | | | | | |
| | L | L | | | |
| 34. I have felt hopeless about the future. | | | | | |
| iuture. | | | | | |
| 35. I have worried that I am a | 1 | [] | | | |
| burden to other people. | | | | | |
| | I | | | | <u> </u> |
| 36. I have wondered why I keep | | | | 100 | |
| going. | | | Walter 17 | | |
| <ol> <li>I have felt angry because of<br/>the disease.</li> </ol> | | | | | |
| ••• | | | | - | |
| 38. I have felt depressed. | | | [] | [ | |
| • | | And the second | | | |
| 39. I have worried about how the | | | | | |
| disease will affect me in the future. | | | | | |
| 40. I have felt as if I have no | | | | | |
| freedom. | | | | | |
| | | | 1 1 | 1 1 | |

Thank you for completing the questionnaire

#### APPENDIX 5 COLUMBIA-SUICIDE SEVERITY RATING SCALE (EXAMPLE)

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Since Last Visit

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide History Form</u>, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc.

| SUICIDAL IDEATION | | | |
|---|---|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suicidal Behavior" section. If the answer to question 2 is "yes", ask questions 3, 4 and 5. If the answer to question 1 and/or 2 is "yes", complete "Intensity of Ideation" section below. | | | |
| 1. Wish to be Dead Subject endorses thoughts about a wish to be dead or not alive anymore, or wish to fall askeep and not wake up. Have you wished you were dead or wished you could go to sleep and not wake up? | | | |
| If yes, describe: | | | |
| 2. Non-Specific Active Suicidal Thoughts General, non-specific thoughts of wanting to end one's life/commit suici oneself/associated methods, intent, or plan during the assessment period. Have you actually had any thoughts of killing yourself? | de (e.g., "I've thought about killing myzelf") without thoughts of ways to kill | Yes | No |
| If yes, describe: | | | |
| 3. Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act Subject endorses thoughts of suicide and has thought of at least one method during the assessment period. This is different than a specific plan with time, place or method details worked out (e.g., thought of method to kill self but not a specific plan). Includes person who would say. "I thought about taking an or erdose but I never made a specific plan as to when, where or how I would actually do itand I would never go through with it." Have you been thinking about how you might do this? | | | |
| If yes, describe: | | | |
| 4. Active Suicidal Ideation with Some Intent to Act, without Specific Plan Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? | | | |
| If yes, describe: | | | |
| 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? | | | |
| If yes, describe: | | | |
| INTENSITY OF IDEATION | | | |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). | | | |
| Most Severe Ideation: Type # (1-5) | Description of Ideation | 1.50 | vere |
| Frequency: How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day | | | |
| Duration When you have the thoughts, how long do they last? | | ŀ | |
| (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time | (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous | | |
| Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty (4) Can control thoughts with little difficulty (5) Unable to control thoughts (6) Can control thoughts with some difficulty (7) Does not strempt to control thoughts | | _ | |
| Deterrents Are there things - anyone or anything (e.g., family, religion thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you | (4) Deterrents the stopped you from wanting to die or acting on (5) Deterrents definitely did not stop you (6) Does not apply | - | |
| Reasons for Ideation What sort of reasons did you have for thinking about wanti | ing to die or killing yourself? Was it to end the pain or stop the way with this pain or how you were feeling) or was it to get attention, (4) Mostly to end or stop the pain (you couldn't go on hving with the pain or how you were feeling) (5) Completely to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (0) Does not apply | _ | _ |

| | <u> </u> | Ŧ |
|---|---|---|
| SUICIDAL BEHAVIOR | Since<br>Vi | |
| (Check all that apply, so long as these are separate events; must ask about all types) Actual Attempt: | | |
| A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as method to kill oneself. Intent | Yes | No |
| does not have to be 100%. If there is all intent desire to die associated with the act, then it can be considered an actual suicide attempt. There does not | | |
| have to be any injury or harm, just the potential for injury or harm. If person pulls trigger while gun is in mouth but gun is broken so no injury results, this is considered an attempt. | | |
| Inferring Intent: Even if an individual denies intent wish to die, it may be inferred clinically from the behavior or circumstances. For example, a highly | | |
| lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from window of a high floor/story). Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be inferred. | | |
| Have you made a strictide attempt? | | |
| Have you done anything to have yourself? | Total | # <b>~</b> £ |
| Have you done anything dangerous where you could have died? | Atter | |
| What did you do? Did you as a way to end your life? | | _ |
| Did you want to die (even a little) when you? | | |
| Were you trying to end your life when you? | | |
| Or did you think it was possible you could have died from | | |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) | | |
| Sympathy, or get sometiming ease to mappeny: (sear-injunous neutral with white state and the control of the con | | |
| | Yes | No |
| Her subject angoged in Non Suigidal Salf Injurious Behavior? | | |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | |
| Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have | Yes | No |
| occurred). | | |
| Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger. | | |
| even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around | | |
| neck but has not yet started to hang - is stopped from doing so. Has there been a time when you started to do something to end your life but someone or something stopped you before you | Total | |
| actually did anything? | intern | upted |
| If yes, describe: | _ | |
| Aborted Attempt: When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. | Yes | No |
| Examples are similar to interrupted attempts, except that the individual stops him herself, instead of being stopped by something else. | | |
| Has there been a time when you started to do something to try to end your life but you stopped yourself before you | Total | # of |
| actually did anything? If yes, describe: | | ned |
| Preparatory Acts or Behavior: | | · |
| Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a | Yes | No _ |
| specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, | | |
| giving valuables away or writing a suicide note)? | | |
| If yes, describe: | | |
| Suicidal Behavior: | Yes | No |
| Suicidal behavior: Suicidal behavior was present during the assessment period? | | |
| Smicide: | Yes | No |
| June | | |
| Assure for Astrol Attended Only | Most Le | |
| Answer for Actual Attempts Only | Attempt | |
| Actual Lethality/Medical Damage: | Date:<br>Enter | Cada |
| O. No physical damage or very minor physical damage (e.g., surface scratches). | Enter | COM |
| 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding, sprains). | | |
| Moderate physical damage: medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns.) | | |
| less than 20% of body; extensive blood loss but can recover, major fractures). | — | |
| 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). | | |
| 5. Desth | 1 | |
| Potential Lethality: Only Answer if Actual Lethality=0 | Enter | Code |
| Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality, put gun in mouth and pulled the trigger but gun fails to fire so no medical damage, laying on train tracks with oncoming train but pulled away. | | |
| perous unit over). | | |
| 0 = Behavior not likely to result in injury | | |
| 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite svailable medical care | | |

Posner K, Brent D, Lucas C, et al. Columbia-Suicide Severity Rating Scale. Version 1/14/09. Standardized Evaluation in Clinical Practice, pp. 103 -130, 200.